CLINICAL TRIAL: NCT02092467
Title: PHASE 3B/4 RANDOMIZED SAFETY ENDPOINT STUDY OF 2 DOSES OF TOFACITINIB IN COMPARISON TO A TUMOR NECROSIS FACTOR (TNF) INHIBITOR IN SUBJECTS WITH RHEUMATOID ARTHRITIS
Brief Title: Safety Study Of Tofacitinib Versus Tumor Necrosis Factor (TNF) Inhibitor In Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3921133; 2013-003177-99 (EudraCT Number)
Record Dates: First submitted 2014-03-03; First posted 2014-03-20 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Arthritis, Rheumatoid
Keywords: Post-marketing; Phase 4; Open-label; Safety Surveillance; CP690550; Xeljanz; oral treatment
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Adalimumab; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment Arm 1 (Experimental)
  Interventions: Drug: tofacitinib
- Treatment Arm 2 (Experimental)
  Interventions: Drug: tofacitinib
- Treatment Arm 3 (Active Comparator): TNF inhibitor Arm - adalimumab will be used in US, Canada and Puerto Rico; etanercept will be used in all other countries.
  Interventions: Biological: adalimumab; Biological: etanercept

INTERVENTIONS:
Drug: tofacitinib — Oral tablet, 5 mg BID
  Arms: Treatment Arm 1
Drug: tofacitinib — Oral tablet, 10 mg BID
  Arms: Treatment Arm 2
Biological: adalimumab — Pre-filled syringe, 40 mg subcutaneous injection, every other week
  Other Names: Humira
  Arms: Treatment Arm 3
Biological: etanercept — Pre-filled syringe, 50 mg subcutaneous injection, every week
  Other Names: Enbrel
  Arms: Treatment Arm 3

SUMMARY:
This post-marketing study is designed to compare the safety of tofacitinib versus TNF inhibitor with respect to major cardiovascular adverse events and malignancies, excluding non-melanoma skin cancers when given to subjects with rheumatoid arthritis. Other safety events, including non-melanoma skin cancers, hepatic events, infections, and efficacy parameters will be collected and evaluated in the study.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe rheumatoid arthritis
* Taking methotrexate without adequate control of symptoms
* Have at least one cardiovascular risk factor (eg, current smoker, high blood pressure, high cholesterol levels, diabetes mellitus, history of heart attack, family history of coronary heart disease, extra-articular RA disease)

Exclusion Criteria:

* Current or recent infection
* Clinically significant laboratory abnormalities
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4372 (Actual)
Dates: Start 2014-03-14 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (344):
- United States (141):
  - University of Alabama at Birmingham (UAB), Arthritis Clinical Intervention Program, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Clinical and Translational Research Center of Alabama, PC, Tuscaloosa, Alabama
  - Southern Arizona VA Health Care System (SAVAHCS), Tucson, Arizona
  - University of Arizona Clinical and Translational Science Research Center, Tucson, Arizona
  - CHI St. Vincent Medical Group Hot Springs, Hot Springs, Arkansas
  - Arthritis And Rheumatism Associates LLC, Jonesboro, Arkansas
  - Medvin Clinical Research, Covina, California
  - Med Investigations, Inc., Fair Oaks, California
  - Talbert Medical Group, Huntington Beach, California
  - University of California, San Diego (UCSD)- Perlman Ambulatory Clinic, La Jolla, California
  - Valerius Medical Group And Research Center Of Greater Long Beach, Inc., Long Beach, California
  - ProHealth Partners, Long Beach, California
  - Keck Medicine of USC, Los Angeles, California
  - California Medical Research Associates Inc, Northridge, California
  - Desert Medical Advances, Palm Desert, California
  - Medvin Clinical Research, Placentia, California
  - Sierra Rheumatology, Inc., Roseville, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Dr. Orrin M. Troum, Md And Medical Associates, Santa Monica, California
  - Los Angeles Biomedical Research Institute at Harbor UCLA Medical Center, Torrance, California
  - Harbor UCLA Medical Center, Torrance, California
  - Robin K. Dore M.D., Inc., Tustin, California
  - Medvin Clinical Research, Van Nuys, California
  - Ventura Clinical Trials, Ventura, California
  - Desert Valley Medical Group, Victorville, California
  - Medvin Clinical Research, Whittier, California
  - Arthritis Associates and Osteoporosis Center of Colorado Springs, Colorado Springs, Colorado
  - Howard University Hospital, Washington D.C., District of Columbia
  - RASF-Clinical Research Center, Inc, Boca Raton, Florida
  - Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - Arthritis & Rheumatism Associates (Private Practice), Clearwater, Florida
  - Florida Clinical Research Group (Administrative Office), Clearwater, Florida
  - Dr.Robert W. Levin MDOffice of, Clearwater, Florida
  - International Medical Research, Daytona Beach, Florida
  - Centre for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - University of Florida - Rheumatology at ACC, Jacksonville, Florida
  - University of Florida College of Medicine, Jacksonville - Rheumatology Research, Jacksonville, Florida
  - Doctors Research Institute, Miami, Florida
  - Center for Arthritis and Rheumatic Diseases, Miami, Florida
  - San Marcus Research Clinic, Miami Lakes, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Advanced Clinical Research of Orlando, Ocoee, Florida
  - Arthritis & osteoporosis treatment center,PA, Orange Park, Florida
  - Rheumatology Associates of Central Florida, PA, Orlando, Florida
  - Omega Research Consultants, LLC, Orlando, Florida
  - Millennium Research, Ormond Beach, Florida
  - Arthritis Center, Inc., Palm Harbor, Florida
  - Arthritis Research of Florida, Inc., Palm Harbor, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Advanced Urgent Care, Port Orange, Florida
  - USF Health Morsani Center for Advanced Healthcare, Tampa, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Arthritis and Rheumatology of GA, P.C., Atlanta, Georgia
  - Medical Associates of North Georgia - Rheumatology, Canton, Georgia
  - Office of Jefrey D. Lieberman, MD, PC, Decatur, Georgia
  - Coeur D'Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - Quincy Medical Group, Quincy, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Diagnostic Rheumatology and Research PC, Indianapolis, Indiana
  - MidWest Clinical Research, LLC, Overland Park, Kansas
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Arthritis and Diabetes Clinic, Inc., Monroe, Louisiana
  - Klein & Associates, M.D.,P.A., Cumberland, Maryland
  - Arthritis Treatment Center, Frederick, Maryland
  - Klein & Associates, MD, PA, Hagerstown, Maryland
  - The Center for Rheumatology and Bone Research, a division of Arthritis and Rheumatism Associates, PC, Wheaton, Maryland
  - Phase III Clinical Research, Fall River, Massachusetts
  - UMass Memorial Medical Center, Memorial Campus, Worcester, Massachusetts
  - Bronson Healthcare Group, Battle Creek, Michigan
  - Bronson Rheumatology Specialists, Kalamazoo, Michigan
  - Jasper Clinic, Inc., Kalamazoo, Michigan
  - Western Michigan University Homer Stryker M.D. School of Medicine Center for Clinical Research, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Borgess Research Institute, Kalamazoo, Michigan
  - June DO,PC, Lansing, Michigan
  - Shores Rheumatology P.C., Saint Clair Shores, Michigan
  - St. Paul Rheumatology, PA, Eagan, Minnesota
  - Center for Diagnostic Imaging, Mendota Heights, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City Internal Medicine, Kansas City, Missouri
  - Clinvest Research, LLC, Springfield, Missouri
  - Glacier View Research Institute, Kalispell, Montana
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Westroads Clinical Research, Inc., Omaha, Nebraska
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Steinberg Diagnostics, Las Vegas, Nevada
  - EKSAKTI, LLC (dba: Eksakti Clinical Research), Las Vegas, Nevada
  - Arthritis Center Of Reno, Reno, Nevada
  - Nashua Rheumatology, Nashua, New Hampshire
  - Summit Medical Group, Clifton, New Jersey
  - Weill Cornell Physicians at Brooklyn Heights, Brooklyn, New York
  - Northwell Health Division of Rheumatology, Great Neck, New York
  - NYU Langone Rheumatology Associates Long Island., Lake Success, New York
  - EmergeOrtho,P.A., Durham, North Carolina
  - Physicians East, PA, Greenville, North Carolina
  - PMG Research of Hickory LLC, Hickory, North Carolina
  - Frycare outpatient imaging Center, Hickory, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - PMG Research Inc., d/b/a PMG Research of Piedmont HealthCare, Statesville, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Trinity Health Center - Medical Arts, Minot, North Dakota
  - Cincinnati Rheumatic Disease Study Group, Inc., Cincinnati, Ohio
  - STAT Research, Inc., Dayton, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Medical Research Foundation (OMRF), Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - The Arthritis Group, Philadelphia, Pennsylvania
  - UPMC Arthritis and Autoimmunity Clinic, Pittsburgh, Pennsylvania
  - UPMC Lupus Center of Excellence, Pittsburgh, Pennsylvania
  - Clinical Research Center of Reading, LLC, Wyomissing, Pennsylvania
  - Rheumatology Associates, P.A., Charleston, South Carolina
  - Innovative Clinical Research, LLC, Greenville, South Carolina
  - Piedmont Arthritis Clinic, PA, Greenville, South Carolina
  - Articluaris Healthcare Group d/b/a ACME Research, Orangeburg, South Carolina
  - Articularis Healthcare Group, Inc d/b/a Low Country Rheumatology, Summerville, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Rheumatology Consultants, PLLC, Knoxville, Tennessee
  - Dr. Ramesh C. Gupta MD, Office of, Memphis, Tennessee
  - Center For Inflammatory Disease, Nashville, Tennessee
  - Amarillo Center for Clinical Research, Ltd., Amarillo, Texas
  - Austin Regional Clinic, Austin, Texas
  - Trinity Universal Research Associates, Inc, Carrollton, Texas
  - Pioneer Research Solutions, Inc., Cypress, Texas
  - Baylor Scott and White Research Institute / Arthritis Care and Research Center, Dallas, Texas
  - Arthritis Centers of Texas, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Accurate Clinical Management, LLC, Houston, Texas
  - Rheumatic Disease Clinical Research Center, Houston, Texas
  - Accurate Clinical Research, Inc., Houston, Texas
  - Houston Institute for Clinical Research, Houston, Texas
  - Medical Center Research, LLC, Houston, Texas
  - Accurate Clinical Research, Inc., League City, Texas
  - Arthritis and Osteoporosis Associates, LLP, Lubbock, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - Trinity Universal Research Associates, Inc., Plano, Texas
  - Center for Arthritis and Rheumatic Diseases, PC, Chesapeake, Virginia
  - Center for Arthritis and Rheumatic Diseases, P.C., Suffolk, Virginia
  - Rheumatic Disease Center, Glendale, Wisconsin
- Argentina (11):
  - OMI- Organizacion Medica de Investigacion, Buenos Aires, Buenos Aires F.D.
  - Centro de Educacion Medica e Investigaciones Clinicas Norberto Quirno (CEMIC), C.a.b.a., Buenos Aires F.D.
  - Sanatorio Parque S.A y Consultorios Externos Asociados, Rosario, Santa Fe Province
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Consultorios Reumatologicos Pampa., Buenos Aires
  - CIER - Centro de Investigaciones en Enfermedades Reumaticas, CABA
  - Centro Privado de Medicina Familiar - Mindout Research S.R.L., CABA
  - Hospital Privado Centro Medico de Cordoba S.A., Córdoba
  - Sanatorio Parque S.A y Consultorios Externos Asociados, Rosario
  - I.A.R.I. Instituto de Asistencia Reumatologica Integral - Sede IMAC, San Isidro
  - CER San Juan, San Juan
- Australia (5):
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - St. Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - Austin Repatriation Hospital, Heidelberg, Victoria
  - Austin Health - Repatriation Hospital, Heidelberg West, Victoria
  - RK Will Pty Ltd, Victoria Park, Western Australia
- Brazil (16):
  - CEDOES - Centro de Diagnostico e Pesquisa da Osteoporose do Espirito Santo, Vitória, Espírito Santo
  - SER - Servicos Especializados em Reumatologia da Bahia, Salvador, Estado de Bahia
  - Hospital das Clinicas Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - CMIP- Centro Mineiro de Pesquisa Ltda/CETAL- Centro de Estudos e Tratamento do Aparelho Locomotor, Juiz de Fora, Minas Gerais
  - EDUMED - Educacao em Saude SS Ltda, Curitiba, Paraná
  - CCBR Brasil - Centro de Pesquisas e Analises Clinicas LTDA, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clinicas de Porto Alegre - UFRGS, Porto Alegre, Rio Grande do Sul
  - Clinica Medica Bonfliglioli Ltda., Campinas, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São Jose Do Rio Preto, São Paulo
  - CPCLin - Centro de Pesquisas Clinicas Ltda. / Clinica Dr. Freddy Goldberg Eliaschewitz LTDA EPP, São Paulo, São Paulo
  - AACD- Lar Escola\ Associacao de Assistencia a Crianca Deficiente, São Paulo, São Paulo
  - Instituto de Assistencia Medica do Hospital do Servidor Publico Estadual, São Paulo, São Paulo
  - Fundacao Faculdade de Medicina MECMPAS - Hospital das Clinicas da FMUSP, São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
  - Hospital Moinhos de Vento, Rio Grande de Sul
  - CEPIC - Centro Paulista de Investigacao Clinica e Servicos Medicos Ltda, São Paulo
- Bulgaria (5):
  - UMBAL "Dr Georgi Stranski" EAD, Pleven
  - MBAL Eurohospital Plovdiv OOD, Plovdiv
  - MBAL RUSe AD,, Rousse
  - UMBAL Sveti Ivan Rilski" EAD, Sofia
  - MBAL Sveta Marina EAD, Varna
- Canada (6):
  - Rheumatology Research Associates, Edmonton, Alberta
  - PerCuro Clinical Research Limited, Victoria, British Columbia
  - Medicine Professional Corporation, Ottawa, Ontario
  - Clinical Research and Arthritis Centre, Windsor, Ontario
  - Centre de Rhumatologie de l'Est du Quebec, Rimouski, Quebec
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
- Chile (3):
  - Centro Medico de Reumatologia Ltda., Temuco, Región de la Araucanía
  - Prosalud, Santiago, Santiago Metropolitan
  - Centro de Investigacion Clinica Universidad Catolica (CICUC), Santiago, Santiago Metropolitan
- Guangdong General Hospital, Guangzhou, Guangdong, China
- Colombia (5):
  - Centro Integral de Reumatologia REUMALAB S.A.S., Medellín, Antioquia
  - Centro de Investigacion en Reumatologia y Especialidades Medicas S.A.S, CIREEM S.A.S, Bogota D.C., Cundinamarca
  - Centro de Investigaciones Clinica del Country, Bogota, Cundinamarca
  - Preventive Care S.A.S., Chía, Cundinamarca
  - Servimed S.A.S, Bucaramanga, Santander Department
- Czechia (9):
  - Vesalion, s.r.o., Ostrava, Czech Republic
  - Mediscan Group, s.r.o., Prague, Czech Republic
  - REVMACLINIC s.r.o., Brno
  - Revmatologie, s.r.o., Brno
  - Revmacentrum MUDr. Mostera, s.r.o., Brno-Židenice
  - Artroscan, s.r.o., Ostrava
  - Revmatologicky ustav., Prague
  - Revmatologicka Ambulance, Prague
  - PV - MEDICAL s.r.o., Zlín
- Finland (3):
  - Helsingin yliopistollinen keskussairaala, Helsinki
  - Kiljavan Laaketutkimus Oy, Hyvinkää
  - Laakarikeskus Aava Hyvinkaan Pipetti, Hyvinkää
- Hong Kong (4):
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan, HKG
  - The University of Hong Kong (HKU)-Queen Mary Hospital (QMH), Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- Israel (10):
  - Barzilai Medical Center - Rheumatology Outpatient Clinic, Ashkelon
  - Assaf Harofeh Medical Center, Beer Yaacov
  - Bnai Zion Medical Center Rheumatology Unit, Haifa
  - Rambam Health Care Campus, Haifa
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center - Hebrew University Hospital, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Jordan (2):
  - Istishari Hospital, Amman
  - King Abdullah University Hospital, Irbid
- Lebanon (2):
  - Hotel Dieu de France Hospital, El Achrafiyé, Beyrouth
  - Ain Wazein Hospital, Lebanon
- Malaysia (3):
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Selayang, Department of Medicine, Batu Caves, Selangor
- Mexico (13):
  - Unidad de Enfermedades Reumaticas y Cronico Degenerativas S. C., Torreón, Coahuila
  - Centro Integral en Reumatologia SA de CV, Guadalajara, Jalisco
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Consultorio de Reumatologia, Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Centro de Investigacion Clinica de Morelia. S.C, Morelia, Michoacán
  - Clinica de Enfermedades Cronicas y Procedimientos Especiales, SC, Morelia, Michoacán
  - Centro de Investigacion de Tratamientos Innovadores de Sinaloa, S.C, Culiacán, Sinaloa
  - Unidad Reumatologica Las Americas S.C.P., Mérida, Yucatán
  - Investigacion y Biomedicina de Chihuahua SC, Chihuahua City
  - CINTRE, Centro de Investigacion y Tratamiento Reumatologico S.C., Mexico City
  - Centro de Alta Especialidad en Reumatologia e Investigacion del Potosi, S.C., San Luis Potosí City
  - Unidad de Investigaciones Reumatologicas, San Luis Potosí City
- Netherlands (2):
  - Medical Center Leeuwarden, Leeuwarden
  - Universitair Medisch Centrum (UMC) Utrecht, Utrecht
- New Zealand (4):
  - Middlemore Hospital Middlemore Clinical Trials Trust, Auckland
  - Rheumatology Clinic, Waikato Hospital, Hamilton
  - Timaru Hospital, Timaru
  - Wellington Hospital, Wellington
- Peru (10):
  - Centro de Investigacion Clinica Trujillo E.I.R.L. Clinica Peruana Americana, Trujillo, La Libertad
  - Centro de lnvestigacion de la Red Asistencial del Hospital Nacional ESSALUD Carlos Alberto Seguin E., Arequipa
  - ACQ MEDIC S.A.C. - Centro de Investigacion Clinica Inmunoreumatologia, Lima
  - Unidad de Investigacion de la Clinica Internacional - Clinica Internacional, Lima
  - ABK REUMA S.R.L. de Medicentro Biociencias- BIO CIENCIAS PERU S.R.L., Lima
  - Instituto Peruano del Hueso y la Articulacion - Instituto Peruano del Hueso y la Articulacion S.A.C., Lima
  - Investigaciones en Reumatologia - Centro Medico Corpac, Lima
  - Investigaciones Clinicas S.A.C., Lima
  - Centro de Investigacion de Reumatologia - Clinica San Borja, Lima
  - Centro de Investigacion en Salud - Centro de Excelencia en Reumatologia, Lima
- Poland (18):
  - NZOZ Lecznica MAK-MED, Nadarzyn, Masovian Voivodeship
  - Zdrowie Osteo-Medic s.c. Lidia i Artur Racewicz, Agnieszka i Jerzy Supronik, Bialystok, Podlaskie Voivodeship
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Kliniczno-Badawcze J.Brzezicki, B.Gornikiewicz-Brzezicka Lekarze Spolka Partnerska, Elblag
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - Centrum Medyczne Pratia Katowice, Katowice
  - Indywidualna Praktyka lekarska Dr hab. med. Anna Szczepańska - Szerej, Lublin
  - Zespol Poradni Specjalistycznych Reumed Filia Onyksowa, Lublin
  - PROFMEDICUS Sp. z o.o., Osrodek Badan Klinicznych, Olsztyn
  - Prywatna Praktyka Lekarska Prof. UM dr hab. med. Pawel Hrycaj, Poznan
  - Pomorskie Centrum Reumatologiczne im. Dr Jadwigi Titz-Kosko w Sopocie, Spolka. z o.o., Sopot
  - KO-MED Centra Kliniczne Sp. zo.o., Staszów
  - NASZ LEKARZ Przychodnie Medyczne, Torun
  - Centrum Medyczne Pratia Warszawa, Warsaw
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - Synexus Polska Sp. z o.o., Wroclaw
  - NZOZ Biogenes Sp. z o.o., Wroclaw
- Puerto Rico (2):
  - Ponce Medical School Foundation, Inc., Ponce
  - Fundacion de Investigaction de Diego, San Juan
- Russia (11):
  - Saint-Petersburg State Budgetary Institution of Healthcare Municipal hospital # 40 of the, Saint Petersburg, St.petersburg
  - SBHI City Clinical Hospital #4 of HD of Moscow, Moscow
  - SBHI of Moscow City Clinical Hospital 1 n. a. N.I. Pirogov of the Healthcare Department of Moscow, Moscow
  - SBIH of Nizhniy Novgorod region City Clinical Hospital #5 of Nizhniy Novgorod district, Nizhny Novgorod
  - Federal State Budgetary Scientific Institution "Research Institute of Fundamental and, Novosibirsk
  - Consulting and Diagnostic Rheumatological Center Healthy Joints LLC, Novosibirsk
  - GBUZ RK Republic Hospital n. a. V.A. Baranov of the MoH & social development Of The Karelia Republic, Petrozavodsk
  - Saint-Petersburg State Budget Healthcare Institution Consultative-diagnostic Center #85, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education, Smolensk
  - SBEI of HPE Ural State Medical University of the MoH of the RF, Yekaterinburg
  - Municipal Budgetary Institution "Central City Clinical Hospital #6", Yekaterinburg
- Slovakia (7):
  - Nestatna reumatologicka ambulancia, Bratislava
  - ROMJAN s.r. o. , Specializovana Reumatologicka ambulancia, Bratislava - Petrzalka
  - AAGS, s.r.o., Reumatologicka ambulancia, Dunajská Streda
  - ECCLESIA s.r.o, Reumatologicka ambulancia, Nové Zámky
  - REUMACENTRUM s.r.o., Reumatologicka ambulancia, Partizánske
  - Reumex s.r.o, Rimavská Sobota
  - Reuma-Global s.r.o., Reumatologicka ambulancia, Trnava
- South Africa (11):
  - Greenacres Hospital, Port Elizabeth, Eastern Cape
  - Wits Clinical Research Site, Johannesburg, Gauteng
  - Clinresco Centres ( Pty ) Ltd, Kempton Park, Gauteng
  - Jakaranda Hospital, Pretoria, Gauteng
  - Emmed Research, Pretoria, Gauteng
  - St. Augustine's Hospital - Chelmsford Medical Centre 2, Durban, KwaZulu-Natal
  - Tiervlei Trial Centre, Karl Bremer Hospital, Bellville, Cape Town, Western Cape
  - Arthritis Clinical Research Trials cc, Cape Town, Western Cape
  - Panorama Medical Centre, Cape Town, Western Cape
  - University of Cape Town, Cape Town, Western Cape
  - Winelands Medical Research Centre-, Stellenbosch
- Spain (10):
  - Hospital de Merida, Mérida, Badajoz
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Nuestra Senora de la Esperanza, Santiago de Compostela, LA Coruna
  - Hospital Universitario de Cruces, Barakaldo, Vizcaya
  - Hospital Universitario de Basurto, Bilbao, Vizcaya
  - Hospital Plato, Barcelona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen de la Macarena, Seville
- Taiwan (7):
  - China Medical University Hospital, Taichung, Taiwan (r.o.c)
  - Changhua Christian Hospital, Changhua
  - Buddhist Dalin Tzu Chi General Hospital, Chiayi City
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou Branch, Taoyuan
- Thailand (5):
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi Hospital, Mahidol University, Bangkok
  - Faculty of Medicine , Siriraj Hospital , Mahidol University, Bangkok
  - Division of Rheumatology, Department of Internal Medicine, Faculty of Medicine,Chiang Mai University, Chiang Mai
  - Prince of Songkla University, Songkhla
- Turkey (Türkiye) (9):
  - Ankara Universitesi Tip Fakultesi Ibn-i Sina Hastanesi, Ankara
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Adnan Menderes Universitesi Tip Fakultesi Hastanesi, Aydin
  - Gaziantep Universitesi Tip Fakultesi, Gaziantep
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Izmir Tepecik Egitim ve Arastirma Hastanesi, Izmir
  - Kocaeli Universitesi Tip Fakultesi Hastanesi, Kocaeli
  - Ondokuz Mayis Universitesi Tip Fakultesi Fiziksel Tip ve, Samsun
  - Cumhuriyet Universitesi Tip Fakultesi Hastanesi, Sivas
- United Kingdom (9):
  - Poole Hospital, University Hospitals Dorset NHS Foundation Trust, Poole, Dorset
  - Barking, Havering and Redbridge University Hospitals NHS Trust, Goodmayes, Essex
  - The Royal Wolverhampton NHS Trust-Cannock Chase Hospital, Cannock
  - Aintree University Hospital, Liverpool University Hospitals, Liverpool
  - Clinical trials, Pharmacy Department, Aintree University Hospitals, Liverpool
  - University of Liverpool Academic Rheumatology Unit. Aintree University Hospital. Liverpool Universit, Liverpool
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Clinical Research Facility, Newcastle upon Tyne
  - Northumbria Healthcare NHS Foundation Trust, North Shields
  - Pharmacy Department, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Giles JT, Charles-Schoeman C, Buch MH, Dougados M, Szekanecz Z, Mikuls TR, Ytterberg SR, Koch GG, Kwok K, Cadatal MJ, Menon S, Chen Y, Diehl AM, Rivas JL, Yndestad A, Bhatt DL. Use of statins and its association with major adverse cardiovascular events with tofacitinib vs TNF inhibitors in patients with rheumatoid arthritis with and without atherosclerotic cardiovascular disease. Ann Rheum Dis. 2026 Jan;85(1):103-113. doi: 10.1016/j.ard.2025.08.028. Epub 2025 Sep 23. PMID 40992967
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Batko B, Jeka S, Wiland P, Zielinska A, Stopinska-Polaszewska M, Stajszczyk M, Kosydar-Piechna M, Cadatal MJ, Rivas JL. Geographical Differences in the Safety and Efficacy of Tofacitinib Versus TNFi: A Post Hoc Analysis of ORAL Surveillance. Rheumatol Ther. 2024 Oct;11(5):1217-1235. doi: 10.1007/s40744-024-00693-y. Epub 2024 Jul 26. PMID 39060905
- [Derived] Citera G, Mysler E, Kakehasi AM, Pascual-Ramos V, Masson W, Cadatal MJ, Rivas JL, Sheibanie F, Helling C, Ponce de Leon D. Cardiovascular Events, Malignancies, and Efficacy Outcomes in Latin American Patients With Rheumatoid Arthritis Receiving Tofacitinib or Tumor Necrosis Factor Inhibitors: A Post Hoc Analysis of the ORAL Surveillance Study. J Clin Rheumatol. 2024 Aug 1;30(5):208-216. doi: 10.1097/RHU.0000000000002106. Epub 2024 Jun 17. PMID 38880956
- [Derived] Buch MH, Bhatt DL, Charles-Schoeman C, Giles JT, Mikuls T, Koch GG, Ytterberg S, Nagy E, Jo H, Kwok K, Connell CA, Masri KR, Yndestad A. Risk of extended major adverse cardiovascular event endpoints with tofacitinib versus TNF inhibitors in patients with rheumatoid arthritis: a post hoc analysis of a phase 3b/4 randomised safety study. RMD Open. 2024 Apr 12;10(2):e003912. doi: 10.1136/rmdopen-2023-003912. PMID 38609322
- [Derived] Karpouzas GA, Szekanecz Z, Baecklund E, Mikuls TR, Bhatt DL, Wang C, Sawyerr GA, Chen Y, Menon S, Connell CA, Ytterberg SR, Mortezavi M. Rheumatoid arthritis disease activity and adverse events in patients receiving tofacitinib or tumor necrosis factor inhibitors: a post hoc analysis of ORAL Surveillance. Ther Adv Musculoskelet Dis. 2023 Nov 6;15:1759720X231201047. doi: 10.1177/1759720X231201047. eCollection 2023. PMID 37942277
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Weitz JI, Szekanecz Z, Charles-Schoeman C, Vranic I, Sahin B, Paciga SA, Wang Z, Hyde C, Martin DA. Biomarkers to predict risk of venous thromboembolism in patients with rheumatoid arthritis receiving tofacitinib or tumour necrosis factor inhibitors. RMD Open. 2022 Nov;8(2):e002571. doi: 10.1136/rmdopen-2022-002571. PMID 36323490
- [Derived] Charles-Schoeman C, Buch MH, Dougados M, Bhatt DL, Giles JT, Ytterberg SR, Koch GG, Vranic I, Wu J, Wang C, Kwok K, Menon S, Rivas JL, Yndestad A, Connell CA, Szekanecz Z. Risk of major adverse cardiovascular events with tofacitinib versus tumour necrosis factor inhibitors in patients with rheumatoid arthritis with or without a history of atherosclerotic cardiovascular disease: a post hoc analysis from ORAL Surveillance. Ann Rheum Dis. 2023 Jan;82(1):119-129. doi: 10.1136/ard-2022-222259. Epub 2022 Sep 22. PMID 36137735
- [Derived] Balanescu AR, Citera G, Pascual-Ramos V, Bhatt DL, Connell CA, Gold D, Chen AS, Sawyerr G, Shapiro AB, Pope JE, Schulze-Koops H. Infections in patients with rheumatoid arthritis receiving tofacitinib versus tumour necrosis factor inhibitors: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2022 Nov;81(11):1491-1503. doi: 10.1136/ard-2022-222405. Epub 2022 Aug 3. PMID 35922124
- [Derived] Ytterberg SR, Bhatt DL, Mikuls TR, Koch GG, Fleischmann R, Rivas JL, Germino R, Menon S, Sun Y, Wang C, Shapiro AB, Kanik KS, Connell CA; ORAL Surveillance Investigators. Cardiovascular and Cancer Risk with Tofacitinib in Rheumatoid Arthritis. N Engl J Med. 2022 Jan 27;386(4):316-326. doi: 10.1056/NEJMoa2109927. PMID 35081280
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921133&StudyName=Safety%20Study%20Of%20tofacitinib%20Versus%20Tumor%20Necrosis%20Factor%20%28TNF%29%20Inhibitor%20In%20Subjects%20With%20Rheumatoid%20Arthritis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study started from 14 March 2014 and completed on 22 July 2020.
Groups:
- Tofacitinib 5 mg BID: Participants received tofacitinib 5 milligram (mg) oral tablet twice daily (BID) up to 72 months. Participants were followed up for at least 28 days after last dose of study drug.
- Tofacitinib 10 mg BID: Participants received tofacitinib 10 mg oral tablets (two tablets of 5 mg each) BID up to 72 months. Dose was reduced to tofacitinib 5 mg BID on or after 19 February 2019 as per Study Protocol Amendment 8. Participants were followed up for at least 28 days after last dose of study drug.
- TNFi: In the United States (US), Puerto Rico and Canada, participants randomized to tumor necrosis factor inhibitor (TNFi) arm received adalimumab 40 mg every other week (QOW) by subcutaneous (SC) injection and in all other countries, participants randomized to TNFi arm received etanercept 50 mg once weekly by SC injection up to 72 months. Participants were followed up for at least 28 days after last dose of study drug.
Period: Overall Study
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Started | 1457 | 1457 | 1458
Treated | 1455 | 1456 | 1451
Completed | 1053 | 998 | 1060
Not Completed | 404 | 459 | 398
Not completed — Death | 49 | 66 | 38
Not completed — Lost to Follow-up | 38 | 35 | 40
Not completed — Global Deterioration of Health Status | 1 | 0 | 0
Not completed — Other | 32 | 30 | 24
Not completed — Withdrawal by Subject | 282 | 327 | 289
Not completed — Randomized but not treated | 2 | 1 | 7

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included all participants who were randomized in the study and received at least one dose of the randomized investigational drug (tofacitinib or TNFi).
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi | Total
Number analyzed (Participants) | 1455 | 1456 | 1451 | 4362
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.75 (6.80) | 61.40 (7.07) | 61.30 (7.47) | 61.15 (7.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1169 | 1124 | 1117 | 3410
  Male | 286 | 332 | 334 | 952
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 438 | 482 | 470 | 1390
  Not Hispanic or Latino | 1017 | 974 | 981 | 2972
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 1128 | 1126 | 1099 | 3353
  Race: Black or African American | 63 | 65 | 83 | 211
  Race: Asian | 65 | 56 | 55 | 176
  Race: Other | 199 | 209 | 214 | 622

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Adjudicated Malignancies Excluding Non-melanoma Skin Cancers (NMSC)
Description: Incidence rate (number of participants with event per 100 participant year [PY]) was defined as the total number of participants with admissible events divided by the total (for all qualifying participants) time at risk for the cohort/treatment group of interest. Malignancy events, excluding NMSC were adjudicated by a steering committee. The risk period (RP) was the last contact date. The last contact date was the maximum of (AE start date, AE stop date, last study visit date, withdrawal date, telephone contact date). If a participant died, last contact date was the death date. First events were counted within the RP. If a participant did not have an event or had an event but outside the risk period, the participant was censored at the end of RP.
Time Frame: Baseline up to last contact date (maximum up to 72 months)
Population: SAS included all participants who were randomized in the study and received at least one dose of the randomized investigational drug (tofacitinib or TNFi).
Measure: Number (95% Confidence Interval); unit: participants with event/100 PY
Groups:
- All Tofacitinib: All participants who received treatment in either tofacitinib 5 mg or tofacitinib 10 mg group BID up to 72 months. Participants were followed up for at least 28 days after last dose of study drug.
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | All Tofacitinib | TNFi
Number analyzed (Participants) | 1455 | 1456 | 2911 | 1451
participants with event/100 PY | 1.13 [0.87 to 1.45] | 1.13 [0.86 to 1.45] | 1.13 [0.94 to 1.35] | 0.77 [0.55 to 1.04]
Statistical Analysis 1: Comparison: All Tofacitinib vs TNFi; All Tofacitinib versus TNFi; Test type: Non-Inferiority — Hazard ratio (95% CI) was based on a univariate Cox proportional hazard model with treatment [All Tofacitinib (ie, tofacitinib 5 mg BID and tofacitinib 10 mg BID combined) and TNFi] as covariate; Hazard Ratio (HR) = 1.48, 95% CI 2-sided [1.04 to 2.09] — Primary comparison. Non-inferiority was to be claimed between All Tofacitinib and TNFi if the upper limit of the 95% CI for HR was < 1.8 (non-inferiority criterion)
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Tofacitinib 10 mg BID versus Tofacitinib 5 mg BID; Test type: Non-Inferiority — Hazard ratio (95% CI) was based on a univariate cox proportional hazard model with treatment (tofacitinib 5 mg BID, tofacitinib 10 mg BID and TNFi) as covariate; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.70 to 1.43] — Secondary comparison. Non-inferiority was to be claimed between tofacitinib 10 mg BID and tofacitinib 5 mg BID if the upper limit of the 95% CI for HR was < 2.0 (non-inferiority criterion)
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs TNFi; Tofacitinib 5 mg BID versus TNFi; Test type: Other — [test comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 1.47, 95% CI 2-sided [1.00 to 2.18] — Supportive analysis to the primary comparison between All Tofacitinib vs TNFi
Statistical Analysis 4: Comparison: Tofacitinib 10 mg BID vs TNFi; Tofacitinib 10 mg BID versus TNFi; Test type: Other — [test comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 1.48, 95% CI 2-sided [1.00 to 2.19] — Supportive analysis to the primary comparison between All Tofacitinib vs TNFi

2. Primary Outcome: Incidence Rate of Adjudicated Major Adverse Cardiovascular Events (MACE)
Description: MACE included the cardiovascular death, non-fatal myocardial infarction (MI) and non-fatal stroke of any classification, including reversible focal neurologic defects with imaging evidence of a new cerebral lesion consistent with ischemia or hemorrhage. Incidence rate was defined as the total number of participants with admissible events divided by the total (for all qualifying participants) time at risk for the cohort/treatment group of interest. The risk period (RP) was the minimum of last contact date or last study treatment dose date + 60 days. The last contact date was the maximum of (AE start date, AE stop date, last study visit date, withdrawal date, telephone contact date). If a participant died, last contact date was the death date. First events were counted within the RP. If a participant did not have an event or had an event but outside the risk period, the participant was censored at the end of RP.
Time Frame: Baseline up to last contact date (maximum up to 72 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: participants with event/100 PY
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | All Tofacitinib | TNFi
Number analyzed (Participants) | 1455 | 1456 | 2911 | 1451
participants with event/100 PY | 0.91 [0.67 to 1.21] | 1.05 [0.78 to 1.38] | 0.98 [0.79 to 1.19] | 0.73 [0.52 to 1.01]
Statistical Analysis 1: Comparison: All Tofacitinib vs TNFi; All Tofacitinib versus TNFi; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.91 to 1.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Tofacitinib 10 mg BID versus Tofacitinib 5 mg BID; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.77 to 1.71] — Secondary Comparison. Non-inferiority was to be claimed between tofacitinib 10 mg BID and tofacitinib 5 mg BID if the upper limit of the 95% CI for HR was <2.0 (non-inferiority criterion)
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs TNFi; Tofacitinib 5 mg BID versus TNFi; Test type: Other — [test comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.81 to 1.91] — Supportive analysis to the primary comparison between All Tofacitinib vs TNFi
Statistical Analysis 4: Comparison: Tofacitinib 10 mg BID vs TNFi; Tofacitinib 10 mg BID versus TNFi; Test type: Other — [test comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.94 to 2.18] — Supportive analysis to the primary comparison between All Tofacitinib vs TNFi

3. Secondary Outcome: Incidence Rate of Non-fatal Stroke
Description: Non-fatal stroke included reversible focal neurologic defects with imaging evidence of a new cerebral lesion consistent with ischemia or hemorrhage. Incidence rate was defined as the total number of participants with admissible events divided by the total (for all qualifying participants) time at risk for the cohort/treatment group of interest. The risk period (RP) was the minimum of last contact date or last study treatment dose date + 60 days. The last contact date was the maximum of (AE start date, AE stop date, last study visit date, withdrawal date, telephone contact date). If a participant died, last contact date was the death date. First events were counted within the RP. If a participant did not have an event or had an event but outside the risk period, the participant was censored at the end of RP.
Time Frame: Baseline up to last contact date (maximum up to 72 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: participants with event/100 PY
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
participants with event/100 PY | 0.27 [0.15 to 0.45] | 0.33 [0.19 to 0.53] | 0.34 [0.20 to 0.54]

4. Secondary Outcome: Incidence Rate of Non-fatal Myocardial Infarction
Description: Incidence rate was defined as the total number of participants with admissible events divided by the total (for all qualifying participants) time at risk for the cohort/treatment group of interest. The risk period (RP) was the minimum of last contact date or last study treatment dose date + 60 days. The last contact date was the maximum of (AE start date, AE stop date, last study visit date, withdrawal date, telephone contact date). If a participant died, last contact date was the death date. First events were counted within the RP. If a participant did not have an event or had an event but outside the risk period, the participant was censored at the end of RP.
Time Frame: Baseline up to last contact date (maximum up to 72 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: participants with event/100 PY
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
participants with event/100 PY | 0.37 [0.22 to 0.57] | 0.33 [0.19 to 0.53] | 0.16 [0.07 to 0.31]

5. Secondary Outcome: Incidence Rate of Adjudicated Opportunistic Infection Events Including Tuberculosis
Description: Opportunistic infections (OI) were reviewed and adjudicated by the opportunistic infection review committee (OIRC). Incidence rate was defined as the total number of participants with admissible events divided by the total (for all qualifying participants) time at risk for the cohort/treatment group of interest. The risk period (RP) was the minimum of last contact date or last study treatment dose date + 28 days. The last contact date was the maximum of (AE start date, AE stop date, last study visit date, withdrawal date, telephone contact date). If a participant died, last contact date was the death date. First events were counted within the RP. If a participant did not have an event or had an event but outside the risk period, the participant was censored at the end of RP.
Time Frame: Baseline up to last contact date (maximum up to 72 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: participants with event/100 PY
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
participants with event/100 PY | 0.76 [0.54 to 1.04] | 0.91 [0.66 to 1.22] | 0.42 [0.26 to 0.64]

6. Secondary Outcome: Incidence Rate of Adjudicated Hepatic Events
Description: Hepatic events (adjudicated) included drug-induced liver injury (DILI) - probable, highly likely and definite, DILI - listed separately, DILI - cases meeting classification and severity, participants with elevations of transaminase levels greater than (>) 1* upper limit of normal (ULN), greater than or equal to (>=) 3*ULN, >=5*ULN (based on laboratory values). Incidence rate was the total number of participants with admissible events divided by total (for all qualifying participants) time at risk for the cohort/treatment group of interest. The risk period (RP) was minimum of The risk period (RP) was the minimum of last contact date or last study treatment dose date + 28 days. Last contact date was maximum of (AE start date, AE stop date, last study visit date, withdrawal date, telephone contact date). In case of death, last contact date was death date. First events counted within RP. Participant did not have an event or had an event outside risk period were censored at end of RP.
Time Frame: Baseline up to last contact date (maximum up to 72 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: participants with event/100 PY
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
participants with event/100 PY | 0.90 [0.66 to 1.20] | 1.51 [1.18 to 1.91] | 0.70 [0.49 to 0.97]

7. Secondary Outcome: Incidence Rate of Adjudicated Cardiovascular Events Other Than Major Adverse Cardiovascular Events (MACE)
Description: Cardiovascular events (adjudicated) were death (coronary and non-coronary), MI, all coronary revascularization, unstable angina, new ischemic heart disease, stroke (fatal and non-fatal), transient ischemic attack (TIA), congestive heart failure (CHF), peripheral arterial vascular disease (PAVD), deep vein thrombosis, pulmonary embolism, arterial embolism, arterial thrombosis. Incidence rate was total number of participants with admissible events divided by total (for all qualifying participants) time at risk for cohort/treatment group of interest. Risk period (RP) was the minimum of last contact date or last study treatment dose date + 28 days. Last contact date was maximum of (AE start date, AE stop date, last study visit date, withdrawal date, telephone contact date). In case of death, last contact date was death date. First events counted within RP. Participant did not have an event or had an event outside risk period were censored at end of RP.
Time Frame: Baseline up to last contact date (maximum up to 72 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: participants with event/100 PY
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
participants with event/100 PY | 1.21 [0.92 to 1.55] | 1.45 [1.13 to 1.83] | 1.05 [0.78 to 1.38]

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE was any untoward medical occurrence post treatment; event need not necessarily had causal relationship with treatment or usage. SAE: any untoward medical occurrence at any dose: resulted in death, life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in congenital anomaly. TEAE: event that occurred for first time during effective duration of treatment and not seen prior to start of treatment or event seen prior to start of treatment but increase in severity during treatment. Risk period (RP) for AE: minimum of last contact date or last study treatment dose date+28 days. RP for SAEs: last contact date. Last contact date was maximum: AE start, AE stop, last study visit, withdrawal and telephone contact. In case of death, last contact was death date. First events counted within RP. Participant did not have event or had event outside risk period were censored at end of RP.
Time Frame: AEs: Baseline up to minimum of last contact date or last study treatment dose date+28 days (maximum up to 72 months); SAEs: Baseline up to minimum of last contact date (maximum up to 72 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
Participants
  AEs | 1333 | 1344 | 1308
  SAEs | 373 | 420 | 339

9. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Parameters
Description: Clinically significant laboratory abnormalities: Hematology: hemoglobin, hematocrit, erythrocytes with primary criteria as less than [<] 0.8* lower limit of normal [LLN]), platelets (<0.5* LLN; >1.75* ULN), leukocytes (<0.6*LLN; >1.5*ULN), lymphocytes, lymphocytes/leukocytes, neutrophils, neutrophils/leukocytes (<0.8*LLN; >1.2*ULN), eosinophils, eosinophils/leukocytes, monocytes, monocytes/leukocytes (>1.2*ULN); urinalysis: urine glucose, urine protein, urine hemoglobin, and leukocyte esterase (>=1); chemistry: bilirubin, indirect bilirubin (>1.5*ULN) aspartate aminotransferase, alanine aminotransferase (>3.0*ULN), creatinine, triglycerides, cholesterol (>1.3*ULN) and HDL cholesterol (<0.8*LLN). Risk period (RP) was minimum of last contact date or last study treatment dose date+28 days. Last contact date was (date of death or maximum of dates: AE start, AE stop, last study visit, withdrawal, telephone contact). Participants without event or event outside RP were censored at end of RP.
Time Frame: Baseline up to last contact date (maximum up to 72 months)
Population: Analysis population included all participants from SAS with an abnormal baseline with at least one observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 919 | 911 | 915
Participants | 238 | 252 | 167

10. Secondary Outcome: Incidence Rate of Adjudicated All-Cause Deaths
Description: All-cause death was defined as the death due to any cause during the course of study. Incidence rate was defined as the total number of participants with admissible events divided by the total (for all qualifying participants) time at risk for the cohort/treatment group of interest. Incidence rate of all-cause deaths (adjudicated by Adjudication Committee) was reported in this outcome measure. The risk period (RP) was the minimum of last contact date or last study treatment dose date + 28 days. The last contact date was the maximum of (AE start date, AE stop date, last study visit date, withdrawal date, telephone contact date). If a participant died, last contact date was the death date. First events were counted within the RP. If a participant did not have an event or had an event but outside the risk period, the participant was censored at the end of RP.
Time Frame: Baseline up to last contact date (maximum up to 72 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: participants with event/100 PY
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
participants with event/100 PY
  Deaths-Total | 0.50 [0.33 to 0.74] | 0.80 [0.57 to 1.09] | 0.34 [0.20 to 0.54]
  Deaths - Infections | 0.08 [0.02 to 0.20] | 0.18 [0.08 to 0.35] | 0.06 [0.01 to 0.17]
  Deaths - Cardiovascular Events | 0.25 [0.13 to 0.43] | 0.41 [0.25 to 0.63] | 0.20 [0.10 to 0.36]
  Deaths - Malignancies | 0.10 [0.03 to 0.23] | 0.00 [0.00 to 0.08] | 0.02 [0.00 to 0.11]
  Deaths - Other Causes | 0.08 [0.02 to 0.20] | 0.21 [0.10 to 0.38] | 0.06 [0.01 to 0.17]

11. Secondary Outcome: Number of Participants With Reasons For Permanent or Temporary Discontinuation of Study Medication
Description: Number of participants who permanent or temporary discontinued study medication due to any AE, treatment related AEs, Coronavirus disease 2019 (COVID 19) related AEs, and herpes zoster were reported. The risk period (RP) was the minimum of last contact date or last study treatment dose date + 28 days. The last contact date was the maximum of (AE start date, AE stop date, last study visit date, withdrawal date, telephone contact date). If a participant died, last contact date was the death date. First events were counted within the RP. If a participant did not have an event or had an event but outside the risk period, the participant was censored at the end of RP.
Time Frame: Baseline up to last contact date (maximum up to 72 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
Participants
  Permanent discontinuation: AE | 210 | 304 | 210
  Temporary discontinuation: AEs | 665 | 736 | 576
  Permanent discontinuation: treatment related AE | 111 | 179 | 114
  Temporary discontinuation: treatment related AE | 407 | 458 | 297
  Permanent discontinuation: COVID-19 Related AEs | 0 | 1 | 0
  Temporary discontinuation: COVID-19 Related AEs | 0 | 1 | 1
  Permanent discontinuation: Herpes Zoster | 6 | 13 | 2
  Temporary discontinuation: Herpes Zoster | 104 | 110 | 33

12. Secondary Outcome: Change From Baseline in Disease Activity Score 28-4 (DAS28-4) C-reactive Protein (CRP) at Month 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60 and 63
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis based on a 28-joint assessment. DAS28-4 (CRP) was calculated from number of painful joints out of 28 joints (TJC28) and number of swollen joints out of 28 joints (SJC28), CRP (milligrams per liter [mg/L]) and patient's global assessment of disease activity (PtGA) on a 100 mm Visual Analog Scale (VAS) (scores ranging from 0 millimeter [mm] [very well] to 100 mm [worst], higher scores indicated worse health condition). Total DAS28-4 (CRP) score range: 0 to 9.4, higher score indicated more disease activity. DAS28-4 (CRP) <= 3.2 indicates low disease activity and > 3.2 to <=5.1 indicates moderate disease activity, >5.1 indicates high disease activity, and DAS28-4 (CRP) < 2.6 indicates remission. DAS28-4 (CRP) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP in mg/L +1) + 0.014*PtGA in mm+ 0.96; ln = natural logarithm, sqrt = square root.
Time Frame: Baseline, Months 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60 and 63
Population: Full Analysis Set (FAS): all participants randomized and received at least one dose of drug. Mixed model for repeated measures used without imputation for missing values. Analyses included data while participants were receiving drug. Only visits with N > 50 participants in each treatment group included in analyses. Number of Participants Analyzed: number of participants included in mixed model for repeated measures. Number Analyzed: number of participants evaluable for each specified time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1409 | 1391 | 1386
units on a scale
  Change at Month 2: number analyzed (Participants) | 1325 | 1301 | 1316
  Change at Month 2 | -2.00 (0.03) | -2.14 (0.03) | -1.89 (0.03)
  Change at Month 3: number analyzed (Participants) | 1367 | 1328 | 1317
  Change at Month 3 | -2.28 (0.03) | -2.42 (0.03) | -2.19 (0.03)
  Change at Month 6: number analyzed (Participants) | 1336 | 1298 | 1294
  Change at Month 6 | -2.50 (0.03) | -2.68 (0.03) | -2.40 (0.03)
  Change at Month 9: number analyzed (Participants) | 1286 | 1246 | 1245
  Change at Month 9 | -2.64 (0.03) | -2.80 (0.03) | -2.54 (0.03)
  Change at Month 12: number analyzed (Participants) | 1254 | 1204 | 1197
  Change at Month 12 | -2.70 (0.03) | -2.85 (0.03) | -2.60 (0.03)
  Change at Month 15: number analyzed (Participants) | 1218 | 1171 | 1174
  Change at Month 15 | -2.78 (0.03) | -2.93 (0.03) | -2.67 (0.03)
  Change at Month 18: number analyzed (Participants) | 1184 | 1121 | 1138
  Change at Month 18 | -2.78 (0.03) | -2.95 (0.03) | -2.76 (0.03)
  Change at Month 21: number analyzed (Participants) | 1169 | 1076 | 1115
  Change at Month 21 | -2.82 (0.03) | -2.97 (0.03) | -2.76 (0.03)
  Change at Month 24: number analyzed (Participants) | 1134 | 1051 | 1097
  Change at Month 24 | -2.82 (0.03) | -2.99 (0.03) | -2.77 (0.03)
  Change at Month 27: number analyzed (Participants) | 1099 | 1015 | 1045
  Change at Month 27 | -2.91 (0.03) | -3.03 (0.03) | -2.81 (0.03)
  Change at Month 30: number analyzed (Participants) | 1073 | 999 | 1039
  Change at Month 30 | -2.92 (0.03) | -3.03 (0.03) | -2.89 (0.03)
  Change at Month 33: number analyzed (Participants) | 1055 | 974 | 1037
  Change at Month 33 | -2.89 (0.03) | -3.03 (0.03) | -2.89 (0.03)
  Change at Month 36: number analyzed (Participants) | 1029 | 951 | 1014
  Change at Month 36 | -2.91 (0.03) | -2.98 (0.03) | -2.88 (0.03)
  Change at Month 39: number analyzed (Participants) | 984 | 888 | 960
  Change at Month 39 | -2.96 (0.03) | -2.97 (0.03) | -2.91 (0.03)
  Change at Month 42: number analyzed (Participants) | 851 | 768 | 831
  Change at Month 42 | -2.95 (0.03) | -3.05 (0.03) | -2.93 (0.03)
  Change at Month 45: number analyzed (Participants) | 710 | 642 | 673
  Change at Month 45 | -2.94 (0.04) | -2.96 (0.04) | -2.97 (0.04)
  Change at Month 48: number analyzed (Participants) | 567 | 506 | 537
  Change at Month 48 | -2.98 (0.04) | -2.99 (0.04) | -2.93 (0.04)
  Change at Month 51: number analyzed (Participants) | 458 | 419 | 414
  Change at Month 51 | -3.00 (0.04) | -2.95 (0.04) | -2.96 (0.04)
  Change at Month 54: number analyzed (Participants) | 363 | 329 | 322
  Change at Month 54 | -2.99 (0.04) | -3.01 (0.05) | -2.99 (0.05)
  Change at Month 57: number analyzed (Participants) | 263 | 240 | 247
  Change at Month 57 | -2.97 (0.05) | -2.93 (0.05) | -3.02 (0.05)
  Change at Month 60: number analyzed (Participants) | 182 | 182 | 166
  Change at Month 60 | -3.09 (0.06) | -2.94 (0.06) | -3.01 (0.06)
  Change at Month 63: number analyzed (Participants) | 106 | 108 | 96
  Change at Month 63 | -3.07 (0.08) | -2.99 (0.07) | -3.05 (0.08)

13. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) Score at Month 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60 and 63
Description: SDAI is the numerical sum of five outcome parameters: TJC and SJC both based on a 28-joint assessment, PtGA and physician's global assessment of health (PhyGA) both assessed on a 0 to 100 mm VAS (higher scores indicate greater affection due to disease activity), and CRP (mg/L). SDAI total score ranges from 0 to 86 with higher score indicating greater disease activity. SDAI <=3.3 indicates disease remission, >3.4 to 11 indicates low disease activity >11 to 26 indicates moderate disease activity, and >26 indicates high disease activity. SDAI = (28TJC) + (28SJC) + PhyGA/10 + PtGA/10 + CRP/10.
Time Frame: Baseline, Month 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60 and 63
Population: FAS: all participants randomized and received at least one dose of drug. Mixed model for repeated measures used without imputation for missing values. Analyses included data while participants were receiving drug. Only visits with N > 50 participants in each treatment group included in analyses. Number of Participants Analyzed: number of participants included in mixed model for repeated measures. Number Analyzed: number of participants evaluable for each specified time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1378 | 1356 | 1346
units on a scale
  Change at Month 2: number analyzed (Participants) | 1272 | 1257 | 1258
  Change at Month 2 | -22.95 (0.33) | -23.84 (0.33) | -22.24 (0.33)
  Change at Month 3: number analyzed (Participants) | 1321 | 1280 | 1273
  Change at Month 3 | -25.73 (0.30) | -26.81 (0.30) | -25.26 (0.30)
  Change at Month 6: number analyzed (Participants) | 1288 | 1245 | 1244
  Change at Month 6 | -27.63 (0.28) | -28.93 (0.28) | -27.21 (0.28)
  Change at Month 9: number analyzed (Participants) | 1244 | 1204 | 1197
  Change at Month 9 | -28.81 (0.28) | -30.07 (0.28) | -28.29 (0.28)
  Change at Month 12: number analyzed (Participants) | 1215 | 1168 | 1143
  Change at Month 12 | -29.56 (0.27) | -30.46 (0.27) | -28.71 (0.27)
  Change at Month 15: number analyzed (Participants) | 1172 | 1128 | 1129
  Change at Month 15 | -30.20 (0.25) | -31.15 (0.26) | -29.30 (0.26)
  Change at Month 18: number analyzed (Participants) | 1149 | 1085 | 1092
  Change at Month 18 | -30.14 (0.26) | -31.29 (0.26) | -30.18 (0.26)
  Change at Month 21: number analyzed (Participants) | 1138 | 1040 | 1072
  Change at Month 21 | -30.42 (0.26) | -31.46 (0.26) | -30.36 (0.26)
  Change at Month 24: number analyzed (Participants) | 1092 | 1010 | 1051
  Change at Month 24 | -30.51 (0.26) | -31.56 (0.26) | -30.33 (0.26)
  Change at month 27: number analyzed (Participants) | 1056 | 979 | 1002
  Change at month 27 | -31.16 (0.25) | -31.85 (0.26) | -30.53 (0.26)
  Change at Month 30: number analyzed (Participants) | 1046 | 970 | 996
  Change at Month 30 | -31.27 (0.25) | -32.02 (0.25) | -31.24 (0.25)
  Change at Month 33: number analyzed (Participants) | 1027 | 947 | 997
  Change at Month 33 | -31.06 (0.26) | -31.91 (0.26) | -31.20 (0.26)
  Change at Month 36: number analyzed (Participants) | 994 | 917 | 978
  Change at Month 36 | -31.26 (0.26) | -31.52 (0.27) | -31.09 (0.26)
  Change at Month 39: number analyzed (Participants) | 954 | 857 | 920
  Change at Month 39 | -31.77 (0.25) | -31.51 (0.26) | -31.36 (0.26)
  Change at Month 42: number analyzed (Participants) | 819 | 733 | 800
  Change at Month 42 | -31.62 (0.27) | -32.09 (0.28) | -31.24 (0.27)
  Change at Month 45: number analyzed (Participants) | 692 | 617 | 646
  Change at Month 45 | -31.27 (0.29) | -31.67 (0.30) | -31.85 (0.30)
  Change at Month 48: number analyzed (Participants) | 547 | 485 | 522
  Change at Month 48 | -31.87 (0.31) | -31.59 (0.32) | -31.68 (0.32)
  Change at Month 51: number analyzed (Participants) | 438 | 406 | 400
  Change at Month 51 | -32.15 (0.33) | -31.52 (0.34) | -31.72 (0.34)
  Change at Month 54: number analyzed (Participants) | 347 | 316 | 314
  Change at Month 54 | -31.91 (0.33) | -32.33 (0.35) | -31.95 (0.35)
  Change at Month 57: number analyzed (Participants) | 253 | 235 | 242
  Change at Month 57 | -31.58 (0.41) | -31.61 (0.42) | -31.98 (0.42)
  Change at Month 60: number analyzed (Participants) | 174 | 179 | 161
  Change at Month 60 | -32.84 (0.46) | -31.57 (0.46) | -32.23 (0.48)
  Change at Month 63: number analyzed (Participants) | 102 | 107 | 95
  Change at Month 63 | -32.27 (0.63) | -32.12 (0.62) | -32.27 (0.66)

14. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Score at Month 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60 and 63
Description: CDAI is the numerical sum of four outcome parameters: TJC and SJC both based on a 28-joint assessment, PtGA and PhyGA both assessed on a 0 to 100 mm VAS (higher scores indicate greater affection due to disease activity). CDAI total score ranges from 0 to 76 with higher score indicating greater disease activity. CDAI <=2.8 indicates disease remission, >2.8 to 10 indicates low disease activity, >10 to 22 indicates moderate disease activity, and >22 indicates high disease activity. CDAI = (28TJC) + (28SJC) + PhyGA/10 + PtGA/10.
Time Frame: Baseline, Month 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60 and 63
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1378 | 1356 | 1348
units on a scale
  Change at Month 2: number analyzed (Participants) | 1272 | 1258 | 1264
  Change at Month 2 | -21.99 (0.32) | -22.84 (0.32) | -21.30 (0.32)
  Change at Month 3: number analyzed (Participants) | 1325 | 1281 | 1276
  Change at Month 3 | -24.76 (0.29) | -25.77 (0.29) | -24.29 (0.30)
  Change at Month 6: number analyzed (Participants) | 1292 | 1246 | 1249
  Change at Month 6 | -26.59 (0.27) | -27.82 (0.28) | -26.21 (0.28)
  Change at Month 9: number analyzed (Participants) | 1245 | 1207 | 1200
  Change at Month 9 | -27.78 (0.27) | -29.03 (0.27) | -27.30 (0.27)
  Change at Month 12: number analyzed (Participants) | 1217 | 1169 | 1146
  Change at Month 12 | -28.52 (0.26) | -29.38 (0.26) | -27.73 (0.26)
  Change at Month 15: number analyzed (Participants) | 1177 | 1129 | 1135
  Change at Month 15 | -29.17 (0.25) | -30.06 (0.25) | -28.38 (0.25)
  Change at Month 18: number analyzed (Participants) | 1152 | 1086 | 1096
  Change at Month 18 | -29.12 (0.25) | -30.21 (0.26) | -29.15 (0.25)
  Change at Month 21: number analyzed (Participants) | 1141 | 1041 | 1075
  Change at Month 21 | -29.45 (0.25) | -30.49 (0.26) | -29.40 (0.25)
  Change at Month 24: number analyzed (Participants) | 1093 | 1013 | 1055
  Change at Month 24 | -29.54 (0.25) | -30.49 (0.26) | -29.39 (0.25)
  Change at Month 27: number analyzed (Participants) | 1058 | 979 | 1011
  Change at Month 27 | -30.16 (0.24) | -30.82 (0.25) | -29.54 (0.25)
  Change at Month 30: number analyzed (Participants) | 1049 | 970 | 1002
  Change at Month 30 | -30.27 (0.24) | -30.99 (0.25) | -30.24 (0.25)
  Change at Month 33: number analyzed (Participants) | 1034 | 951 | 1000
  Change at Month 33 | -30.05 (0.25) | -30.85 (0.25) | -30.23 (0.25)
  Change at Month 36: number analyzed (Participants) | 999 | 920 | 982
  Change at Month 36 | -30.29 (0.25) | -30.50 (0.26) | -30.14 (0.25)
  Change at Month 39: number analyzed (Participants) | 958 | 858 | 923
  Change at Month 39 | -30.78 (0.24) | -30.49 (0.25) | -30.35 (0.25)
  Change at Month 42: number analyzed (Participants) | 820 | 736 | 801
  Change at Month 42 | -30.66 (0.26) | -31.05 (0.27) | -30.25 (0.26)
  Change at Month 45: number analyzed (Participants) | 694 | 618 | 650
  Change at Month 45 | -30.28 (0.28) | -30.68 (0.29) | -30.83 (0.29)
  Change at Month 48: number analyzed (Participants) | 547 | 487 | 522
  Change at Month 48 | -30.85 (0.30) | -30.57 (0.32) | -30.69 (0.31)
  Change at Month 51: number analyzed (Participants) | 440 | 407 | 401
  Change at Month 51 | -31.09 (0.32) | -30.50 (0.33) | -30.74 (0.33)
  Change at Month 54: number analyzed (Participants) | 347 | 317 | 314
  Change at Month 54 | -31.03 (0.32) | -31.38 (0.33) | -31.02 (0.33)
  Change at Month 57: number analyzed (Participants) | 254 | 236 | 242
  Change at Month 57 | -30.62 (0.40) | -30.75 (0.41) | -30.95 (0.41)
  Change at Month 60: number analyzed (Participants) | 175 | 179 | 161
  Change at Month 60 | -31.74 (0.45) | -30.57 (0.45) | -31.31 (0.47)
  Change at Month 63: number analyzed (Participants) | 102 | 107 | 95
  Change at Month 63 | -31.23 (0.58) | -31.08 (0.57) | -31.65 (0.60)

15. Secondary Outcome: Percentage of Participants Who Achieved Observed American College of Rheumatology-European League Against Rheumatism (ACR-EULAR) Boolean Remission Criteria
Description: ACR-EULAR Boolean-based definition of remission participant must satisfy all of the following: TJC28 <=1, SJC28 <=1, CRP <=10 mg/L, PtGA on a 0-100 mm scale, higher scores indicate greater affection due to disease activity.
Time Frame: Month 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69 and 72
Population: FAS included all participants randomized in study and received at least one dose of randomized investigational drug. Analyses included data while participants were receiving the study drug. 'Number Analyzed' signifies number of participants evaluable for each specified time point. Last Observation Carried Forward (LOCF) applied for missing components and composite binary outcome was calculated. The percentages were calculated using numbers of participants evaluable at each visit as denominators.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
percentage of participants
  Month 2: number analyzed (Participants) | 1356 | 1342 | 1368
  Month 2 | 3.83 | 4.99 | 3.22
  Month 3: number analyzed (Participants) | 1432 | 1424 | 1427
  Month 3 | 5.73 | 7.72 | 6.10
  Month 6: number analyzed (Participants) | 1417 | 1398 | 1411
  Month 6 | 9.10 | 10.66 | 7.80
  Month 9: number analyzed (Participants) | 1392 | 1349 | 1384
  Month 9 | 10.85 | 12.60 | 8.96
  Month 12: number analyzed (Participants) | 1372 | 1332 | 1360
  Month 12 | 11.22 | 13.06 | 9.12
  Month 15: number analyzed (Participants) | 1353 | 1311 | 1342
  Month 15 | 12.56 | 15.18 | 10.28
  Month 18: number analyzed (Participants) | 1322 | 1284 | 1316
  Month 18 | 12.10 | 16.04 | 11.78
  Month 21: number analyzed (Participants) | 1302 | 1255 | 1294
  Month 21 | 12.90 | 15.22 | 13.45
  Month 24: number analyzed (Participants) | 1287 | 1226 | 1273
  Month 24 | 13.60 | 15.99 | 13.35
  Month 27: number analyzed (Participants) | 1269 | 1211 | 1255
  Month 27 | 13.24 | 17.59 | 14.82
  Month 30: number analyzed (Participants) | 1248 | 1191 | 1237
  Month 30 | 13.46 | 16.96 | 14.31
  Month 33: number analyzed (Participants) | 1232 | 1177 | 1221
  Month 33 | 13.88 | 15.97 | 14.82
  Month 36: number analyzed (Participants) | 1206 | 1162 | 1211
  Month 36 | 14.51 | 16.18 | 14.53
  Month 39: number analyzed (Participants) | 1183 | 1140 | 1201
  Month 39 | 13.78 | 14.30 | 15.15
  Month 42: number analyzed (Participants) | 1163 | 1110 | 1179
  Month 42 | 14.79 | 15.41 | 15.01
  Month 45: number analyzed (Participants) | 1021 | 970 | 1023
  Month 45 | 14.89 | 15.46 | 15.74
  Month 48: number analyzed (Participants) | 865 | 806 | 839
  Month 48 | 15.14 | 13.90 | 17.28
  Month 51: number analyzed (Participants) | 698 | 671 | 689
  Month 51 | 14.33 | 15.50 | 16.26
  Month 54: number analyzed (Participants) | 564 | 548 | 550
  Month 54 | 14.01 | 16.42 | 16.36
  Month 57: number analyzed (Participants) | 444 | 445 | 431
  Month 57 | 15.54 | 14.16 | 15.08
  Month 60: number analyzed (Participants) | 327 | 330 | 321
  Month 60 | 11.31 | 12.73 | 15.58
  Month 63: number analyzed (Participants) | 221 | 230 | 223
  Month 63 | 11.76 | 16.96 | 15.25
  Month 66: number analyzed (Participants) | 122 | 131 | 122
  Month 66 | 9.02 | 16.79 | 13.11
  Month 69: number analyzed (Participants) | 46 | 46 | 48
  Month 69 | 13.04 | 19.57 | 14.58
  Month 72: number analyzed (Participants) | 12 | 18 | 15
  Month 72 | 8.33 | 22.22 | 13.33

16. Secondary Outcome: Percentage of Participants With Simplified Disease Activity Index (SDAI) Less Than or Equal to (<=) 3.3
Description: SDAI is the numerical sum of five outcome parameters: TJC and SJC both based on a 28-joint assessment, PtGA and PhyGA both assessed on a 0 to 100 mm VAS (higher scores indicate greater affection due to disease activity), and CRP (mg/L). SDAI total score ranges from 0 to 86 with higher score indicating greater disease activity. SDAI <=3.3 indicates disease remission, >3.4 to 11 indicates low disease activity >11 to 26 indicates moderate disease activity, and >26 indicates high disease activity. SDAI = (28TJC) + (28SJC) + PhyGA/10 + PtGA/10 + CRP/10.
Time Frame: Month 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69 and 72
Population: FAS included all participants randomized in the study and received at least one dose of investigational drug. Analyses included the data while the participants were receiving the study drug. Here, 'Number Analyzed' signifies number of participants evaluable for each specified time point. LOCF was applied for missing components, and then composite binary outcome was calculated. The percentages were calculated using the numbers of participants evaluable at each visit as the denominators.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
percentage of participants
  Month 2: number analyzed (Participants) | 1320 | 1308 | 1325
  Month 2 | 4.62 | 7.03 | 4.15
  Month 3: number analyzed (Participants) | 1425 | 1409 | 1416
  Month 3 | 9.19 | 11.14 | 7.84
  Month 6: number analyzed (Participants) | 1414 | 1391 | 1404
  Month 6 | 12.38 | 14.23 | 10.40
  Month 9: number analyzed (Participants) | 1390 | 1349 | 1380
  Month 9 | 15.90 | 17.72 | 12.75
  Month 12: number analyzed (Participants) | 1372 | 1332 | 1358
  Month 12 | 15.89 | 18.69 | 13.92
  Month 15: number analyzed (Participants) | 1353 | 1311 | 1340
  Month 15 | 18.26 | 20.29 | 15.90
  Month 18: number analyzed (Participants) | 1322 | 1284 | 1316
  Month 18 | 18.68 | 21.96 | 16.79
  Month 21: number analyzed (Participants) | 1302 | 1255 | 1294
  Month 21 | 20.89 | 22.07 | 17.93
  Month 24: number analyzed (Participants) | 1287 | 1226 | 1273
  Month 24 | 20.44 | 22.76 | 18.93
  Month 27: number analyzed (Participants) | 1269 | 1211 | 1255
  Month 27 | 21.91 | 23.62 | 21.12
  Month 30: number analyzed (Participants) | 1248 | 1191 | 1237
  Month 30 | 21.31 | 23.68 | 21.91
  Month 33: number analyzed (Participants) | 1232 | 1177 | 1221
  Month 33 | 21.43 | 25.06 | 22.19
  Month 36: number analyzed (Participants) | 1206 | 1162 | 1211
  Month 36 | 22.47 | 24.35 | 21.80
  Month 39: number analyzed (Participants) | 1183 | 1140 | 1201
  Month 39 | 22.99 | 24.21 | 21.48
  Month 42: number analyzed (Participants) | 1163 | 1110 | 1179
  Month 42 | 24.59 | 24.23 | 23.41
  Month 45: number analyzed (Participants) | 1021 | 970 | 1023
  Month 45 | 25.27 | 23.20 | 23.26
  Month 48: number analyzed (Participants) | 865 | 806 | 839
  Month 48 | 25.32 | 23.20 | 24.20
  Month 51: number analyzed (Participants) | 698 | 671 | 689
  Month 51 | 23.35 | 23.85 | 24.24
  Month 54: number analyzed (Participants) | 564 | 548 | 550
  Month 54 | 22.34 | 24.09 | 24.55
  Month 57: number analyzed (Participants) | 444 | 445 | 431
  Month 57 | 24.10 | 23.82 | 24.83
  Month 60: number analyzed (Participants) | 327 | 330 | 321
  Month 60 | 18.65 | 20.30 | 25.23
  Month 63: number analyzed (Participants) | 221 | 230 | 223
  Month 63 | 19.00 | 23.48 | 23.32
  Month 66: number analyzed (Participants) | 122 | 131 | 122
  Month 66 | 14.75 | 21.37 | 20.49
  Month 69: number analyzed (Participants) | 46 | 46 | 48
  Month 69 | 17.39 | 17.39 | 22.92
  Month 72: number analyzed (Participants) | 12 | 18 | 15
  Month 72 | 16.67 | 22.22 | 13.33

17. Secondary Outcome: Percentage of Participants With Clinical Disease Activity Index (CDAI) <=2.8
Description: as for outcome 14
Time Frame: Month 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69 and 72
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
percentage of participants
  Month 2: number analyzed (Participants) | 1320 | 1311 | 1330
  Month 2 | 4.70 | 7.40 | 4.36
  Month 3: number analyzed (Participants) | 1425 | 1410 | 1417
  Month 3 | 9.26 | 11.06 | 7.76
  Month 6: number analyzed (Participants) | 1414 | 1391 | 1405
  Month 6 | 12.87 | 14.31 | 10.32
  Month 9: number analyzed (Participants) | 1390 | 1349 | 1381
  Month 9 | 15.76 | 18.09 | 13.25
  Month 12: number analyzed (Participants) | 1372 | 1332 | 1359
  Month 12 | 16.33 | 18.62 | 14.64
  Month 15: number analyzed (Participants) | 1353 | 1311 | 1341
  Month 15 | 18.03 | 21.36 | 16.41
  Month 18: number analyzed (Participants) | 1322 | 1284 | 1316
  Month 18 | 19.82 | 22.12 | 17.93
  Month 21: number analyzed (Participants) | 1302 | 1255 | 1294
  Month 21 | 21.35 | 22.55 | 18.70
  Month 24: number analyzed (Participants) | 1287 | 1226 | 1273
  Month 24 | 20.44 | 22.76 | 19.48
  Month 27: number analyzed (Participants) | 1269 | 1211 | 1255
  Month 27 | 22.77 | 23.29 | 21.51
  Month 30: number analyzed (Participants) | 1248 | 1191 | 1237
  Month 30 | 21.88 | 24.18 | 22.31
  Month 33: number analyzed (Participants) | 1232 | 1177 | 1221
  Month 33 | 22.24 | 25.91 | 22.36
  Month 36: number analyzed (Participants) | 1206 | 1162 | 1211
  Month 36 | 23.22 | 25.30 | 21.64
  Month 39: number analyzed (Participants) | 1183 | 1140 | 1201
  Month 39 | 23.92 | 24.30 | 21.90
  Month 42: number analyzed (Participants) | 1163 | 1110 | 1179
  Month 42 | 25.02 | 24.95 | 23.66
  Month 45: number analyzed (Participants) | 1021 | 970 | 1023
  Month 45 | 25.95 | 24.23 | 23.85
  Month 48: number analyzed (Participants) | 865 | 806 | 839
  Month 48 | 25.55 | 24.44 | 24.31
  Month 51: number analyzed (Participants) | 698 | 671 | 689
  Month 51 | 24.50 | 24.89 | 25.11
  Month 54: number analyzed (Participants) | 564 | 548 | 550
  Month 54 | 23.23 | 25.00 | 25.45
  Month 57: number analyzed (Participants) | 444 | 445 | 431
  Month 57 | 24.32 | 24.04 | 25.75
  Month 60: number analyzed (Participants) | 327 | 330 | 321
  Month 60 | 19.88 | 20.91 | 26.48
  Month 63: number analyzed (Participants) | 221 | 230 | 223
  Month 63 | 20.81 | 22.17 | 22.87
  Month 66: number analyzed (Participants) | 122 | 131 | 122
  Month 66 | 13.93 | 22.14 | 17.21
  Month 69: number analyzed (Participants) | 46 | 46 | 48
  Month 69 | 19.57 | 19.57 | 18.75
  Month 72: number analyzed (Participants) | 12 | 18 | 15
  Month 72 | 16.67 | 22.22 | 13.33

18. Secondary Outcome: Percentage of Participants With Simplified Disease Activity Index (SDAI) <=11
Description: as for outcome 16
Time Frame: Month 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69 and 72
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
percentage of participants
  Month 2: number analyzed (Participants) | 1320 | 1308 | 1325
  Month 2 | 30.76 | 35.02 | 28.08
  Month 3: number analyzed (Participants) | 1425 | 1409 | 1416
  Month 3 | 41.47 | 45.00 | 37.99
  Month 6: number analyzed (Participants) | 1414 | 1391 | 1404
  Month 6 | 50.85 | 53.56 | 45.80
  Month 9: number analyzed (Participants) | 1390 | 1349 | 1380
  Month 9 | 56.40 | 59.82 | 52.90
  Month 12: number analyzed (Participants) | 1372 | 1332 | 1358
  Month 12 | 57.87 | 61.11 | 54.93
  Month 15: number analyzed (Participants) | 1353 | 1311 | 1340
  Month 15 | 61.12 | 63.92 | 57.39
  Month 18: number analyzed (Participants) | 1322 | 1284 | 1316
  Month 18 | 62.10 | 65.19 | 60.41
  Month 21: number analyzed (Participants) | 1302 | 1255 | 1294
  Month 21 | 62.75 | 65.26 | 61.21
  Month 24: number analyzed (Participants) | 1287 | 1226 | 1273
  Month 24 | 63.17 | 66.15 | 61.59
  Month 27: number analyzed (Participants) | 1269 | 1211 | 1255
  Month 27 | 65.17 | 66.97 | 63.67
  Month 30: number analyzed (Participants) | 1248 | 1191 | 1237
  Month 30 | 67.23 | 68.35 | 65.64
  Month 33: number analyzed (Participants) | 1232 | 1177 | 1221
  Month 33 | 65.75 | 68.82 | 65.36
  Month 36: number analyzed (Participants) | 1206 | 1162 | 1211
  Month 36 | 67.33 | 66.61 | 65.48
  Month 39: number analyzed (Participants) | 1183 | 1140 | 1201
  Month 39 | 69.74 | 67.11 | 66.03
  Month 42: number analyzed (Participants) | 1163 | 1110 | 1179
  Month 42 | 68.96 | 70.72 | 66.41
  Month 45: number analyzed (Participants) | 1021 | 970 | 1023
  Month 45 | 68.36 | 68.97 | 67.55
  Month 48: number analyzed (Participants) | 865 | 806 | 839
  Month 48 | 67.28 | 64.76 | 67.94
  Month 51: number analyzed (Participants) | 698 | 671 | 689
  Month 51 | 67.91 | 67.51 | 67.78
  Month 54: number analyzed (Participants) | 564 | 548 | 550
  Month 54 | 64.89 | 68.61 | 68.00
  Month 57: number analyzed (Participants) | 444 | 445 | 431
  Month 57 | 63.51 | 66.29 | 68.21
  Month 60: number analyzed (Participants) | 327 | 330 | 321
  Month 60 | 63.30 | 66.67 | 64.17
  Month 63: number analyzed (Participants) | 221 | 230 | 223
  Month 63 | 61.54 | 68.26 | 64.57
  Month 66: number analyzed (Participants) | 122 | 131 | 122
  Month 66 | 59.02 | 71.76 | 59.02
  Month 69: number analyzed (Participants) | 46 | 46 | 48
  Month 69 | 60.87 | 65.22 | 68.75
  Month 72: number analyzed (Participants) | 12 | 18 | 15
  Month 72 | 50.00 | 66.67 | 60.00

19. Secondary Outcome: Percentage of Participants With Clinical Disease Activity Index (CDAI) <=10
Description: as for outcome 14
Time Frame: Month 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69 and 72
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
percentage of participants
  Month 2: number analyzed (Participants) | 1320 | 1311 | 1330
  Month 2 | 29.47 | 34.25 | 26.92
  Month 3: number analyzed (Participants) | 1425 | 1410 | 1417
  Month 3 | 40.07 | 43.90 | 35.99
  Month 6: number analyzed (Participants) | 1414 | 1391 | 1405
  Month 6 | 49.36 | 51.83 | 43.63
  Month 9: number analyzed (Participants) | 1390 | 1349 | 1381
  Month 9 | 55.40 | 58.78 | 50.91
  Month 12: number analyzed (Participants) | 1372 | 1332 | 1359
  Month 12 | 56.56 | 59.38 | 53.57
  Month 15: number analyzed (Participants) | 1353 | 1311 | 1341
  Month 15 | 60.31 | 62.70 | 55.93
  Month 18: number analyzed (Participants) | 1322 | 1284 | 1316
  Month 18 | 60.51 | 64.02 | 59.42
  Month 21: number analyzed (Participants) | 1302 | 1255 | 1294
  Month 21 | 61.37 | 64.94 | 60.20
  Month 24: number analyzed (Participants) | 1287 | 1226 | 1273
  Month 24 | 62.78 | 65.25 | 61.19
  Month 27: number analyzed (Participants) | 1269 | 1211 | 1255
  Month 27 | 64.93 | 66.39 | 62.87
  Month 30: number analyzed (Participants) | 1248 | 1191 | 1237
  Month 30 | 67.15 | 67.84 | 65.00
  Month 33: number analyzed (Participants) | 1232 | 1177 | 1221
  Month 33 | 65.50 | 67.71 | 65.03
  Month 36: number analyzed (Participants) | 1206 | 1162 | 1211
  Month 36 | 66.67 | 65.15 | 64.66
  Month 39: number analyzed (Participants) | 1183 | 1140 | 1201
  Month 39 | 68.64 | 66.40 | 65.61
  Month 42: number analyzed (Participants) | 1163 | 1110 | 1179
  Month 42 | 68.44 | 69.10 | 65.82
  Month 45: number analyzed (Participants) | 1021 | 970 | 1023
  Month 45 | 67.97 | 68.66 | 67.16
  Month 48: number analyzed (Participants) | 865 | 806 | 839
  Month 48 | 66.71 | 63.15 | 67.58
  Month 51: number analyzed (Participants) | 698 | 671 | 689
  Month 51 | 67.77 | 65.87 | 67.63
  Month 54: number analyzed (Participants) | 564 | 548 | 550
  Month 54 | 64.54 | 67.88 | 68.00
  Month 57: number analyzed (Participants) | 444 | 445 | 431
  Month 57 | 62.61 | 65.39 | 67.98
  Month 60: number analyzed (Participants) | 327 | 330 | 321
  Month 60 | 63.00 | 65.15 | 65.42
  Month 63: number analyzed (Participants) | 221 | 230 | 223
  Month 63 | 62.90 | 66.52 | 66.37
  Month 66: number analyzed (Participants) | 122 | 131 | 122
  Month 66 | 57.38 | 67.94 | 61.48
  Month 69: number analyzed (Participants) | 46 | 46 | 48
  Month 69 | 58.70 | 65.22 | 66.67
  Month 72: number analyzed (Participants) | 12 | 18 | 15
  Month 72 | 50.00 | 66.67 | 53.33

20. Secondary Outcome: Percentage of Participants With Disease Activity Score 28-4 (DAS28-4) C-reactive Protein (CRP) <=3.2
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis based on a 28-joint assessment. DAS28-4 (CRP) was calculated from number of painful joints out of 28 joints (TJC28) and number of swollen joints out of 28 joints (SJC28), CRP (mg/L) and PtGA on a 100 mm VAS (VAS: scores ranging from 0 mm [very well] to 100 mm [worst], higher scores indicated worse health condition). Total DAS28-4 (CRP) score range: 0 to 9.4, higher score indicated more disease activity. DAS28-4 (CRP) <= 3.2 indicates low disease activity and > 3.2 to <=5.1 indicates moderate disease activity, >5.1 indicates high disease activity, and DAS28-4 (CRP) < 2.6 indicates remission. DAS28-4 (CRP) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP in mg/L +1) + 0.014*PtGA in mm+ 0.96.
Time Frame: Month 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69 and 72
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
percentage of participants
  Month 2: number analyzed (Participants) | 1347 | 1327 | 1354
  Month 2 | 31.55 | 35.57 | 28.36
  Month 3: number analyzed (Participants) | 1430 | 1418 | 1420
  Month 3 | 41.68 | 46.05 | 37.54
  Month 6: number analyzed (Participants) | 1416 | 1396 | 1406
  Month 6 | 50.28 | 54.87 | 44.88
  Month 9: number analyzed (Participants) | 1392 | 1349 | 1381
  Month 9 | 56.11 | 59.01 | 50.91
  Month 12: number analyzed (Participants) | 1372 | 1332 | 1359
  Month 12 | 57.73 | 60.06 | 53.05
  Month 15: number analyzed (Participants) | 1353 | 1311 | 1341
  Month 15 | 60.38 | 63.54 | 55.03
  Month 18: number analyzed (Participants) | 1322 | 1284 | 1316
  Month 18 | 61.72 | 63.86 | 58.51
  Month 21: number analyzed (Participants) | 1302 | 1255 | 1294
  Month 21 | 62.29 | 63.67 | 59.27
  Month 24: number analyzed (Participants) | 1287 | 1226 | 1273
  Month 24 | 61.93 | 64.11 | 59.78
  Month 27: number analyzed (Participants) | 1269 | 1211 | 1255
  Month 27 | 64.22 | 67.63 | 60.56
  Month 30: number analyzed (Participants) | 1248 | 1191 | 1237
  Month 30 | 64.66 | 65.49 | 63.22
  Month 33: number analyzed (Participants) | 1232 | 1177 | 1221
  Month 33 | 63.80 | 66.02 | 62.82
  Month 36: number analyzed (Participants) | 1206 | 1162 | 1211
  Month 36 | 64.43 | 64.63 | 62.59
  Month 39: number analyzed (Participants) | 1183 | 1140 | 1201
  Month 39 | 65.85 | 65.18 | 63.53
  Month 42: number analyzed (Participants) | 1163 | 1110 | 1179
  Month 42 | 65.43 | 67.93 | 65.31
  Month 45: number analyzed (Participants) | 1021 | 970 | 1023
  Month 45 | 64.74 | 65.77 | 64.52
  Month 48: number analyzed (Participants) | 865 | 806 | 839
  Month 48 | 64.39 | 64.52 | 64.36
  Month 51: number analyzed (Participants) | 698 | 671 | 689
  Month 51 | 65.19 | 66.47 | 65.46
  Month 54: number analyzed (Participants) | 564 | 548 | 550
  Month 54 | 64.18 | 66.24 | 66.55
  Month 57: number analyzed (Participants) | 444 | 445 | 431
  Month 57 | 63.06 | 63.60 | 67.29
  Month 60: number analyzed (Participants) | 327 | 330 | 321
  Month 60 | 62.69 | 64.24 | 65.11
  Month 63: number analyzed (Participants) | 221 | 230 | 223
  Month 63 | 60.18 | 64.35 | 68.61
  Month 66: number analyzed (Participants) | 122 | 131 | 122
  Month 66 | 55.74 | 66.41 | 60.66
  Month 69: number analyzed (Participants) | 46 | 46 | 48
  Month 69 | 58.70 | 56.52 | 70.83
  Month 72: number analyzed (Participants) | 12 | 18 | 15
  Month 72 | 50.00 | 61.11 | 73.33

21. Secondary Outcome: Number of Participants With an American College of Rheumatology 20 Percent (%) (ACR20) Response
Description: ACR20 response is a >= 20% improvement in TJC (28) and SJC (28) and >=20% improvement in 3 of the 5 remaining ACR-core criteria: 1) PGA of arthritis, 2) PtGA of arthritis, 3) participant's assessment of arthritis pain, 4) participant's assessment of functional disability by HAQ-DI, and 5) CRP (mg/L) at each visit. PGA: physician's global assessment of arthritis on VAS, 0 (very well) to 100 mm (worst arthritis), higher scores=worse condition. PtGA: participant's global assessment of arthritis on VAS, 0 mm (very well) to 100 mm (worst arthritis condition), higher scores = worse condition. Participant's assessment of arthritis pain: assessed on VAS, 0 mm (no pain) to 100 mm (most severe pain), higher score = more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (unable to do), higher score=more disability.
Time Frame: Month 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69 and 72
Population: FAS included all participants randomized in the study and received at least one dose of investigational drug. Analyses included the data while the participants were receiving the study drug. Here, 'Number Analyzed' signifies number of participants evaluable for each specified time point. LOCF was applied for missing components, and then composite binary outcome was calculated.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
Participants
  Month 2: number analyzed (Participants) | 1335 | 1316 | 1337
  Month 2 | 832 | 867 | 812
  Month 3: number analyzed (Participants) | 1418 | 1398 | 1396
  Month 3 | 979 | 992 | 923
  Month 6: number analyzed (Participants) | 1402 | 1375 | 1382
  Month 6 | 999 | 1012 | 981
  Month 9: number analyzed (Participants) | 1375 | 1328 | 1356
  Month 9 | 1019 | 1004 | 987
  Month 12: number analyzed (Participants) | 1362 | 1308 | 1333
  Month 12 | 1033 | 992 | 966
  Month 15: number analyzed (Participants) | 1341 | 1291 | 1315
  Month 15 | 1017 | 1003 | 969
  Month 18: number analyzed (Participants) | 1309 | 1266 | 1289
  Month 18 | 981 | 974 | 937
  Month 21: number analyzed (Participants) | 1289 | 1238 | 1271
  Month 21 | 955 | 953 | 949
  Month 24: number analyzed (Participants) | 1275 | 1209 | 1251
  Month 24 | 956 | 922 | 922
  Month 27: number analyzed (Participants) | 1255 | 1190 | 1234
  Month 27 | 961 | 917 | 913
  Month 30: number analyzed (Participants) | 1237 | 1173 | 1213
  Month 30 | 932 | 899 | 931
  Month 33: number analyzed (Participants) | 1220 | 1157 | 1194
  Month 33 | 935 | 888 | 922
  Month 36: number analyzed (Participants) | 1193 | 1145 | 1189
  Month 36 | 907 | 881 | 887
  Month 39: number analyzed (Participants) | 1172 | 1122 | 1180
  Month 39 | 896 | 843 | 887
  Month 42: number analyzed (Participants) | 1153 | 1091 | 1154
  Month 42 | 905 | 848 | 883
  Month 45: number analyzed (Participants) | 1010 | 955 | 1006
  Month 45 | 780 | 718 | 790
  Month 48: number analyzed (Participants) | 854 | 795 | 821
  Month 48 | 654 | 587 | 639
  Month 51: number analyzed (Participants) | 691 | 659 | 675
  Month 51 | 535 | 485 | 518
  Month 54: number analyzed (Participants) | 559 | 536 | 538
  Month 54 | 434 | 396 | 400
  Month 57: number analyzed (Participants) | 441 | 436 | 421
  Month 57 | 337 | 321 | 302
  Month 60: number analyzed (Participants) | 323 | 323 | 314
  Month 60 | 243 | 237 | 232
  Month 63: number analyzed (Participants) | 217 | 221 | 220
  Month 63 | 163 | 166 | 161
  Month 66: number analyzed (Participants) | 119 | 130 | 122
  Month 66 | 85 | 101 | 89
  Month 69: number analyzed (Participants) | 46 | 46 | 48
  Month 69 | 26 | 36 | 37
  Month 72: number analyzed (Participants) | 11 | 18 | 15
  Month 72 | 5 | 15 | 10

22. Secondary Outcome: Number of Participants With an American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response is a >= 50% improvement in TJC (28) and SJC (28) and >=50% improvement in 3 of the 5 remaining ACR-core criteria: 1) PGA of arthritis, 2) PtGA of arthritis, 3) participant's assessment of arthritis pain, 4) participant's assessment of functional disability by HAQ-DI, and 5) CRP (mg/L) at each visit. PGA: physician's global assessment of arthritis on VAS, 0 (very well) to 100 mm (worst arthritis), higher scores=worse condition. PtGA: participant's global assessment of arthritis on VAS, 0 mm (very well) to 100 mm (worst arthritis condition), higher scores = worse condition. Participant's assessment of arthritis pain: assessed on VAS, 0 mm (no pain) to 100 mm (most severe pain), higher score = more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (unable to do), higher score=more disability.
Time Frame: Month 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69 and 72
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
Participants
  Month 2: number analyzed (Participants) | 1337 | 1321 | 1346
  Month 2 | 402 | 452 | 336
  Month 3: number analyzed (Participants) | 1422 | 1405 | 1404
  Month 3 | 528 | 561 | 460
  Month 6: number analyzed (Participants) | 1408 | 1378 | 1387
  Month 6 | 605 | 614 | 533
  Month 9: number analyzed (Participants) | 1381 | 1333 | 1356
  Month 9 | 620 | 651 | 577
  Month 12: number analyzed (Participants) | 1362 | 1312 | 1334
  Month 12 | 631 | 654 | 577
  Month 15: number analyzed (Participants) | 1340 | 1290 | 1313
  Month 15 | 652 | 668 | 582
  Month 18: number analyzed (Participants) | 1312 | 1265 | 1290
  Month 18 | 633 | 643 | 609
  Month 21: number analyzed (Participants) | 1290 | 1234 | 1272
  Month 21 | 607 | 623 | 608
  Month 24: number analyzed (Participants) | 1276 | 1209 | 1249
  Month 24 | 622 | 616 | 592
  Month 27: number analyzed (Participants) | 1258 | 1194 | 1231
  Month 27 | 620 | 602 | 596
  Month 30: number analyzed (Participants) | 1236 | 1177 | 1213
  Month 30 | 599 | 609 | 610
  Month 33: number analyzed (Participants) | 1220 | 1158 | 1200
  Month 33 | 585 | 611 | 594
  Month 36: number analyzed (Participants) | 1195 | 1143 | 1188
  Month 36 | 603 | 566 | 592
  Month 39: number analyzed (Participants) | 1170 | 1121 | 1179
  Month 39 | 595 | 588 | 561
  Month 42: number analyzed (Participants) | 1151 | 1093 | 1161
  Month 42 | 592 | 578 | 587
  Month 45: number analyzed (Participants) | 1011 | 955 | 1008
  Month 45 | 521 | 481 | 519
  Month 48: number analyzed (Participants) | 854 | 794 | 826
  Month 48 | 422 | 385 | 424
  Month 51: number analyzed (Participants) | 693 | 659 | 677
  Month 51 | 350 | 320 | 346
  Month 54: number analyzed (Participants) | 560 | 538 | 540
  Month 54 | 284 | 271 | 268
  Month 57: number analyzed (Participants) | 440 | 437 | 422
  Month 57 | 200 | 210 | 209
  Month 60: number analyzed (Participants) | 325 | 322 | 314
  Month 60 | 152 | 151 | 150
  Month 63: number analyzed (Participants) | 220 | 223 | 219
  Month 63 | 100 | 104 | 103
  Month 66: number analyzed (Participants) | 122 | 129 | 121
  Month 66 | 52 | 68 | 55
  Month 69: number analyzed (Participants) | 45 | 45 | 47
  Month 69 | 16 | 20 | 27
  Month 72: number analyzed (Participants) | 11 | 18 | 15
  Month 72 | 3 | 6 | 7

23. Secondary Outcome: Number of Participants With an American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response is a >= 70% improvement in TJC (28) and SJC (28) and >=70% improvement in 3 of the 5 remaining ACR-core criteria: 1) PGA of arthritis, 2) PtGA of arthritis, 3) participant's assessment of arthritis pain, 4) participant's assessment of functional disability by HAQ-DI, and 5) CRP (mg/L) at each visit. PGA: physician's global assessment of arthritis on VAS, 0 (very well) to 100 mm (worst arthritis), higher scores=worse condition. PtGA: participant's global assessment of arthritis on VAS, 0 mm (very well) to 100 mm (worst arthritis condition), higher scores = worse condition. Participant's assessment of arthritis pain: assessed on VAS, 0 mm (no pain) to 100 mm (most severe pain), higher score = more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (unable to do), higher score=more disability.
Time Frame: Month 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69 and 72
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1455 | 1456 | 1451
Participants
  Month 2: number analyzed (Participants) | 1343 | 1326 | 1354
  Month 2 | 152 | 193 | 113
  Month 3: number analyzed (Participants) | 1425 | 1414 | 1413
  Month 3 | 253 | 268 | 199
  Month 6: number analyzed (Participants) | 1409 | 1388 | 1397
  Month 6 | 282 | 331 | 234
  Month 9: number analyzed (Participants) | 1383 | 1336 | 1366
  Month 9 | 328 | 367 | 291
  Month 12: number analyzed (Participants) | 1364 | 1312 | 1338
  Month 12 | 337 | 373 | 284
  Month 15: number analyzed (Participants) | 1342 | 1294 | 1323
  Month 15 | 359 | 390 | 304
  Month 18: number analyzed (Participants) | 1311 | 1269 | 1295
  Month 18 | 358 | 382 | 325
  Month 21: number analyzed (Participants) | 1293 | 1238 | 1277
  Month 21 | 362 | 370 | 322
  Month 24: number analyzed (Participants) | 1279 | 1211 | 1255
  Month 24 | 349 | 386 | 328
  Month 27: number analyzed (Participants) | 1259 | 1192 | 1238
  Month 27 | 374 | 390 | 342
  Month 30: number analyzed (Participants) | 1238 | 1177 | 1221
  Month 30 | 369 | 397 | 358
  Month 33: number analyzed (Participants) | 1222 | 1160 | 1204
  Month 33 | 357 | 392 | 355
  Month 36: number analyzed (Participants) | 1195 | 1145 | 1193
  Month 36 | 362 | 343 | 351
  Month 39: number analyzed (Participants) | 1173 | 1125 | 1186
  Month 39 | 371 | 361 | 338
  Month 42: number analyzed (Participants) | 1152 | 1098 | 1163
  Month 42 | 376 | 342 | 343
  Month 45: number analyzed (Participants) | 1010 | 957 | 1006
  Month 45 | 313 | 298 | 298
  Month 48: number analyzed (Participants) | 855 | 794 | 826
  Month 48 | 256 | 228 | 238
  Month 51: number analyzed (Participants) | 691 | 657 | 677
  Month 51 | 216 | 195 | 199
  Month 54: number analyzed (Participants) | 559 | 538 | 538
  Month 54 | 159 | 163 | 160
  Month 57: number analyzed (Participants) | 441 | 438 | 421
  Month 57 | 128 | 127 | 118
  Month 60: number analyzed (Participants) | 326 | 321 | 315
  Month 60 | 79 | 83 | 92
  Month 63: number analyzed (Participants) | 220 | 223 | 219
  Month 63 | 58 | 57 | 64
  Month 66: number analyzed (Participants) | 122 | 130 | 122
  Month 66 | 25 | 38 | 35
  Month 69: number analyzed (Participants) | 46 | 45 | 48
  Month 69 | 8 | 15 | 14
  Month 72: number analyzed (Participants) | 11 | 18 | 15
  Month 72 | 2 | 5 | 4

24. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at Months 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60 and 63
Description: HAQ-DI assesses the degree of difficulty a participant has experienced during the past week in 8 domains of daily living activities: dressing/grooming; arising; eating; walking; reach; grip; hygiene; and other activities. There were total of 30 items distributed in these 8 domains. Each item was scored on a 4-point scale from 0 to 3: 0= no difficulty; 1= some difficulty; 2= much difficulty; 3= unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0 (least difficulty) and 3 (extreme difficulty), where higher scores indicate more difficulty while performing daily living activities.
Time Frame: Baseline, Months 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60 and 63
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
Number analyzed (Participants) | 1409 | 1390 | 1388
units on a scale
  Change at Month 2: number analyzed (Participants) | 1325 | 1301 | 1323
  Change at Month 2 | -0.42 (0.02) | -0.45 (0.02) | -0.38 (0.02)
  Change at Month 3: number analyzed (Participants) | 1371 | 1329 | 1320
  Change at Month 3 | -0.45 (0.02) | -0.48 (0.02) | -0.42 (0.02)
  Change at Month 6: number analyzed (Participants) | 1341 | 1297 | 1299
  Change at Month 6 | -0.50 (0.02) | -0.51 (0.02) | -0.46 (0.02)
  Change at Month 9: number analyzed (Participants) | 1287 | 1247 | 1248
  Change at Month 9 | -0.51 (0.02) | -0.55 (0.02) | -0.47 (0.02)
  Change at Month 12: number analyzed (Participants) | 1256 | 1205 | 1200
  Change at Month 12 | -0.52 (0.02) | -0.53 (0.02) | -0.49 (0.02)
  Change at Month 15: number analyzed (Participants) | 1223 | 1171 | 1179
  Change at Month 15 | -0.53 (0.02) | -0.56 (0.02) | -0.51 (0.02)
  Change at Month 18: number analyzed (Participants) | 1189 | 1122 | 1143
  Change at Month 18 | -0.52 (0.02) | -0.56 (0.02) | -0.49 (0.02)
  Change at Month 21: number analyzed (Participants) | 1172 | 1076 | 1118
  Change at Month 21 | -0.53 (0.02) | -0.55 (0.02) | -0.50 (0.02)
  Change at Month 24: number analyzed (Participants) | 1135 | 1052 | 1101
  Change at Month 24 | -0.52 (0.02) | -0.57 (0.02) | -0.49 (0.02)
  Change at Month 27: number analyzed (Participants) | 1102 | 1015 | 1054
  Change at Month 27 | -0.52 (0.02) | -0.56 (0.02) | -0.51 (0.02)
  Change at Month 30: number analyzed (Participants) | 1078 | 998 | 1045
  Change at Month 30 | -0.53 (0.02) | -0.55 (0.02) | -0.50 (0.02)
  Change at Month 33: number analyzed (Participants) | 1063 | 977 | 1041
  Change at Month 33 | -0.51 (0.02) | -0.56 (0.02) | -0.52 (0.02)
  Change at Month 36: number analyzed (Participants) | 1034 | 953 | 1020
  Change at Month 36 | -0.50 (0.02) | -0.54 (0.02) | -0.48 (0.02)
  Change at Month 39: number analyzed (Participants) | 989 | 892 | 964
  Change at Month 39 | -0.51 (0.02) | -0.54 (0.02) | -0.49 (0.02)
  Change at Month 42: number analyzed (Participants) | 854 | 770 | 833
  Change at Month 42 | -0.51 (0.02) | -0.52 (0.02) | -0.50 (0.02)
  Change at Month 45: number analyzed (Participants) | 713 | 642 | 678
  Change at Month 45 | -0.50 (0.02) | -0.51 (0.02) | -0.51 (0.02)
  Change at Month 48: number analyzed (Participants) | 569 | 509 | 539
  Change at Month 48 | -0.50 (0.02) | -0.50 (0.02) | -0.48 (0.02)
  Change at Month 51: number analyzed (Participants) | 461 | 420 | 416
  Change at Month 51 | -0.53 (0.02) | -0.49 (0.02) | -0.50 (0.02)
  Change at Month 54: number analyzed (Participants) | 364 | 330 | 324
  Change at Month 54 | -0.53 (0.02) | -0.51 (0.02) | -0.48 (0.02)
  Change at Month 57: number analyzed (Participants) | 266 | 240 | 247
  Change at Month 57 | -0.49 (0.02) | -0.48 (0.02) | -0.48 (0.02)
  Change at Month 60: number analyzed (Participants) | 185 | 181 | 167
  Change at Month 60 | -0.52 (0.03) | -0.49 (0.03) | -0.48 (0.03)
  Change at Month 63: number analyzed (Participants) | 107 | 108 | 96
  Change at Month 63 | -0.54 (0.03) | -0.48 (0.03) | -0.48 (0.04)

ADVERSE EVENTS:
Time Frame: Baseline up to last contact date (maximum up to 72 months)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. SAS included all participants randomized in the study and received at least one dose of the randomized investigational drug. Total 153 deaths of which 152 were adjudicated and 1 occurred after the participant discontinued from the study.
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | TNFi
All-Cause Mortality (participants affected / at risk) | 49/1455 | 66/1456 | 38/1451
Serious Adverse Events (participants affected / at risk) | 373/1455 | 420/1456 | 339/1451
Other Adverse Events (participants affected / at risk) | 1108/1455 | 1127/1456 | 1056/1451
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 5 mg BID (N=1455) | Tofacitinib 10 mg BID (N=1456) | TNFi (N=1451)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 9 | 4 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Cytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1 | 4
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 4 | 2 | 3
Angina unstable (Cardiac disorders) | 3 | 3 | 3
Aortic valve disease (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 2 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 8 | 6
Atrial flutter (Cardiac disorders) | 2 | 1 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 4 | 0
Cardiac failure (Cardiac disorders) | 2 | 3 | 3
Cardiac failure acute (Cardiac disorders) | 2 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 6 | 0
Cardiac pseudoaneurysm (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 0
Chronic left ventricular failure (Cardiac disorders) | 1 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 2 | 0 | 0
Coronary artery disease (Cardiac disorders) | 8 | 3 | 1
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 2 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 4
Myocardial ischaemia (Cardiac disorders) | 4 | 3 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 3
Right ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 3 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 | 1 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0
Exomphalos (Congenital, familial and genetic disorders) | 0 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 1
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 1
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Adrenal disorder (Endocrine disorders) | 1 | 0 | 0
Adrenal haematoma (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 2
Cataract (Eye disorders) | 3 | 6 | 3
Diabetic retinopathy (Eye disorders) | 0 | 1 | 0
Episcleritis (Eye disorders) | 0 | 0 | 1
Keratoconus (Eye disorders) | 0 | 1 | 0
Macular hole (Eye disorders) | 0 | 1 | 0
Necrotising retinitis (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Retinal vasculitis (Eye disorders) | 0 | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 1 | 0
Uveitis (Eye disorders) | 0 | 1 | 1
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 4 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 1
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 3 | 1 | 2
Gastritis erosive (Gastrointestinal disorders) | 1 | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal erosion (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 4
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 2
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 3 | 3
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Ischaemic enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Jejunal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Jejunal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Obturator hernia (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2 | 2
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 2 | 0
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 2 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3
Accidental death (General disorders) | 1 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 1
Chest discomfort (General disorders) | 3 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 1
Complication associated with device (General disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 2 | 4
Device intolerance (General disorders) | 0 | 1 | 0
Drug intolerance (General disorders) | 0 | 1 | 1
Impaired healing (General disorders) | 0 | 1 | 0
Inflammation (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 1
Non-cardiac chest pain (General disorders) | 4 | 5 | 5
Oedema peripheral (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 3 | 2
Sudden death (General disorders) | 0 | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 2 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 3 | 3
Cholecystitis acute (Hepatobiliary disorders) | 3 | 2 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 2 | 2
Cholelithiasis (Hepatobiliary disorders) | 4 | 5 | 4
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 2
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 1 | 0
Gallbladder rupture (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 2
Hepatorenal failure (Hepatobiliary disorders) | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Abscess (Infections and infestations) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 3 | 1 | 1
Acute pulmonary histoplasmosis (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Adenovirus infection (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 2 | 0 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 4 | 4 | 0
Appendicitis perforated (Infections and infestations) | 2 | 0 | 0
Arthritis bacterial (Infections and infestations) | 2 | 4 | 4
Arthritis infective (Infections and infestations) | 0 | 2 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 2
Bacteraemia (Infections and infestations) | 1 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0
Bone tuberculosis (Infections and infestations) | 0 | 1 | 0
Brain abscess (Infections and infestations) | 1 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 10 | 9 | 7
Bronchitis bacterial (Infections and infestations) | 2 | 0 | 0
Bronchitis viral (Infections and infestations) | 1 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 2
COVID-19 (Infections and infestations) | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 5 | 1
Carbuncle (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 12 | 13 | 15
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 1
Cholecystitis infective (Infections and infestations) | 1 | 1 | 1
Chorioretinitis (Infections and infestations) | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 2 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Colonic abscess (Infections and infestations) | 0 | 1 | 0
Complicated appendicitis (Infections and infestations) | 2 | 0 | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 2 | 2 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 2 | 1
Disseminated varicella zoster virus infection (Infections and infestations) | 0 | 4 | 0
Diverticulitis (Infections and infestations) | 7 | 6 | 2
Encephalitis meningococcal (Infections and infestations) | 0 | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1
Escherichia pyelonephritis (Infections and infestations) | 2 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 2
External ear cellulitis (Infections and infestations) | 0 | 1 | 0
Extradural abscess (Infections and infestations) | 1 | 1 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 4 | 7 | 3
Gastroenteritis bacterial (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 2 | 0
Herpes oesophagitis (Infections and infestations) | 0 | 0 | 1
Herpes ophthalmic (Infections and infestations) | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 9 | 11 | 2
Histoplasmosis (Infections and infestations) | 0 | 1 | 0
Infected bite (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 4 | 3 | 2
Intervertebral discitis (Infections and infestations) | 1 | 0 | 1
Joint abscess (Infections and infestations) | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 3 | 1
Lung abscess (Infections and infestations) | 0 | 1 | 0
Lyme disease (Infections and infestations) | 1 | 0 | 0
Medical device site joint infection (Infections and infestations) | 1 | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 0 | 1
Meningoencephalitis herpetic (Infections and infestations) | 0 | 1 | 0
Muscle abscess (Infections and infestations) | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 1 | 0
Neuroborreliosis (Infections and infestations) | 0 | 0 | 1
Neurocryptococcosis (Infections and infestations) | 1 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 2 | 3 | 1
Osteomyelitis acute (Infections and infestations) | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0
Parotid abscess (Infections and infestations) | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 2 | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 0
Pericarditis tuberculous (Infections and infestations) | 1 | 0 | 0
Perihepatic abscess (Infections and infestations) | 0 | 1 | 0
Peritoneal tuberculosis (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 1 | 1
Pneumonia (Infections and infestations) | 50 | 56 | 43
Pneumonia bacterial (Infections and infestations) | 2 | 1 | 3
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 1
Pneumonia legionella (Infections and infestations) | 1 | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 2 | 1 | 1
Post procedural pneumonia (Infections and infestations) | 0 | 0 | 1
Post procedural sepsis (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 3 | 2 | 2
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 3
Pulpitis dental (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 2 | 2 | 1
Pyelonephritis acute (Infections and infestations) | 2 | 1 | 0
Pyometra (Infections and infestations) | 0 | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 1
Renal abscess (Infections and infestations) | 0 | 0 | 1
Renal tuberculosis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 2 | 2
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 1
Retroperitoneal abscess (Infections and infestations) | 0 | 0 | 1
Salmonella sepsis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 6 | 6 | 5
Septic shock (Infections and infestations) | 4 | 9 | 3
Sinobronchitis (Infections and infestations) | 0 | 0 | 1
Sinusitis fungal (Infections and infestations) | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 1 | 0
Systemic candida (Infections and infestations) | 1 | 0 | 0
Tick-borne fever (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Tubo-ovarian abscess (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 2
Urinary tract infection (Infections and infestations) | 14 | 14 | 9
Urosepsis (Infections and infestations) | 0 | 3 | 2
Viral infection (Infections and infestations) | 1 | 2 | 2
Wound infection (Infections and infestations) | 1 | 1 | 2
Wound infection staphylococcal (Infections and infestations) | 0 | 1 | 0
Wound sepsis (Infections and infestations) | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 5 | 4
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Central cord syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Complicated fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 | 3 | 4
Femur fracture (Injury, poisoning and procedural complications) | 10 | 5 | 11
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 3 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Graft complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 5 | 4 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 5 | 3 | 4
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 3 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 3 | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 3 | 1 | 4
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 4
Skin laceration (Injury, poisoning and procedural complications) | 3 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1 | 4
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subarachnoid haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 3 | 4
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 2 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Biopsy endometrium normal (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 2 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 4 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 2
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone hypertrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Hip deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 29 | 23 | 16
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 11 | 10 | 12
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spinal instability (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Synovial disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Thoracic spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gallbladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Heavy chain disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian granulosa cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1 | 0
Basilar artery stenosis (Nervous system disorders) | 0 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 2
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 1
Cervical cord compression (Nervous system disorders) | 0 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1
Coma hepatic (Nervous system disorders) | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 3
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 2 | 0
Facial paralysis (Nervous system disorders) | 0 | 3 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 4 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Hypoglycaemic seizure (Nervous system disorders) | 1 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 1
Intracranial mass (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 2 | 0 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Morton's neuralgia (Nervous system disorders) | 1 | 0 | 0
Myelopathy (Nervous system disorders) | 2 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0
Postictal paralysis (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Progressive supranuclear palsy (Nervous system disorders) | 0 | 1 | 0
Quadriplegia (Nervous system disorders) | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 3 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 2 | 1 | 0
Seizure (Nervous system disorders) | 2 | 3 | 0
Senile dementia (Nervous system disorders) | 0 | 1 | 0
Spinal claudication (Nervous system disorders) | 1 | 0 | 0
Spondylitic myelopathy (Nervous system disorders) | 1 | 1 | 1
Status epilepticus (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 3 | 5
Thecal sac compression (Nervous system disorders) | 1 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 8 | 4
Vascular encephalopathy (Nervous system disorders) | 0 | 0 | 1
Device dislocation (Product Issues) | 2 | 2 | 2
Device failure (Product Issues) | 2 | 0 | 0
Device loosening (Product Issues) | 0 | 3 | 0
Device occlusion (Product Issues) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 2 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 2
Mental status changes (Psychiatric disorders) | 0 | 3 | 3
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 6 | 2
Bladder diverticulum (Renal and urinary disorders) | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 2 | 0 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 2
Renal atrophy (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 2 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 2 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Renal injury (Renal and urinary disorders) | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 1 | 2
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 2
Cervical polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 | 0 | 0
Endometrial thickening (Reproductive system and breast disorders) | 0 | 1 | 0
Genital prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Orchitis noninfective (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 2 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 22 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 5
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aortic intramural haematoma (Vascular disorders) | 0 | 1 | 0
Aortic occlusion (Vascular disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 2 | 1 | 1
Aortitis (Vascular disorders) | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 7 | 2
Extremity necrosis (Vascular disorders) | 0 | 0 | 1
Femoral artery embolism (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 2 | 3
Hypertensive crisis (Vascular disorders) | 0 | 1 | 2
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1
Hypertensive urgency (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 2
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0
Iliac artery occlusion (Vascular disorders) | 1 | 0 | 0
Labile blood pressure (Vascular disorders) | 0 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 3 | 0 | 2
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
Varicose ulceration (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 3 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 5 mg BID (N=1455) | Tofacitinib 10 mg BID (N=1456) | TNFi (N=1451)
Anaemia (Blood and lymphatic system disorders) | 75 | 100 | 73
Lymphopenia (Blood and lymphatic system disorders) | 107 | 151 | 36
Diarrhoea (Gastrointestinal disorders) | 99 | 81 | 74
Nausea (Gastrointestinal disorders) | 67 | 96 | 61
Bronchitis (Infections and infestations) | 221 | 243 | 168
Gastroenteritis (Infections and infestations) | 61 | 76 | 52
Herpes zoster (Infections and infestations) | 175 | 160 | 59
Influenza (Infections and infestations) | 92 | 95 | 71
Latent tuberculosis (Infections and infestations) | 89 | 72 | 94
Nasopharyngitis (Infections and infestations) | 168 | 172 | 164
Pharyngitis (Infections and infestations) | 87 | 81 | 75
Sinusitis (Infections and infestations) | 97 | 81 | 94
Upper respiratory tract infection (Infections and infestations) | 319 | 318 | 264
Urinary tract infection (Infections and infestations) | 190 | 220 | 186
Fall (Injury, poisoning and procedural complications) | 177 | 160 | 159
Alanine aminotransferase increased (Investigations) | 67 | 75 | 48
Arthralgia (Musculoskeletal and connective tissue disorders) | 111 | 90 | 124
Back pain (Musculoskeletal and connective tissue disorders) | 101 | 113 | 112
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 84 | 71 | 77
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 183 | 188 | 202
Headache (Nervous system disorders) | 50 | 75 | 64
Cough (Respiratory, thoracic and mediastinal disorders) | 77 | 70 | 72
Hypertension (Vascular disorders) | 129 | 152 | 127

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT02092467/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT02092467/SAP_001.pdf